CLINICAL TRIAL: NCT00790933
Title: A Phase 3, Open-label Study to Determine the Long-term Safety and Efficacy of Vedolizumab (MLN0002) in Subjects With Ulcerative Colitis and Crohn's Disease
Brief Title: An Open-label Study of Vedolizumab (MLN0002) in Participants With Ulcerative Colitis and Crohn's Disease
Acronym: GEMINI LTS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: C13008; 2008-002784-14 (EudraCT Number); NMRR-08-1040-2195 (Registry Identifier: NMRR); CTRI/2009/091/000138 (Registry Identifier: CTRI); 10/H1102/12 (Registry Identifier: NRES); NL25209.096.08 (Registry Identifier: CCMO)
Record Dates: First submitted 2008-11-05; First posted 2008-11-14 (Estimated); Results first posted 2019-03-12 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Ulcerative Colitis; Crohn's Disease
Keywords: Drug therapy
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease | interventions — vedolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Vedolizumab 300 mg (Experimental): Vedolizumab 300 mg, 30-minute intravenous (IV) infusion every 4 weeks, starting at Week 0 for approximately up to 510 weeks.
  Interventions: Drug: Vedolizumab

INTERVENTIONS:
Drug: Vedolizumab — Vedolizumab intravenous infusion
  Other Names: MLN0002

SUMMARY:
The purpose of this multicenter, open-label study is to collect data on the occurrence of important clinical safety events resulting from chronic vedolizumab (MLN0002) administration.

DETAILED DESCRIPTION:
The drug being tested in this study is called vedolizumab. Vedolizumab is being tested to treat people who have ulcerative colitis or Crohn's disease. This study will determine the safety profile of long-term vedolizumab treatment.

The study enrolled 2243 patients. Participants who received either placebo or vedolizumab 300 mg IV infusion every 4 or 8 weeks in previous vedolizumab studies received:

• Vedolizumab 300 mg

All participants received vedolizumab intravenous infusion every 4 weeks for approximately up to 510 weeks.

This multicenter trial is being conducted worldwide. The overall time to participate in this study was up to October 2017 until vedolizumab was available in the country in which the participant resided, or until participant withdrawal, whichever came first. Participants made multiple visits to the clinic up to 16 weeks after receiving their last dose of vedolizumab and were being followed up for 2-years during which a safety questionnaire was administered by telephone for follow-up assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Previous treatment in Study C13004 (NCT00619489), Study C13006 (NCT00783718), Study C13007 (NCT00783692), or Study C13011 (NCT01224171) that, in the opinion of the investigator, was well tolerated OR b. Moderate to severe Crohn's disease or ulcerative colitis which has not been previously treated with vedolizumab (MLN0002)
2. May be receiving a therapeutic dose of conventional therapies for Crohn's disease or ulcerative colitis as defined by the protocol

Exclusion Criteria:

1. Development of any new, unstable, or uncontrolled disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2243 (Actual)
Dates: Start 2009-05-22 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2017-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor Clinical Science, Study Director — Takeda
Locations (41):
- United States (31):
  - Birmingham, Alabama
  - San Diego, California
  - San Francisco, California
  - Lafayette, Colorado
  - Littleton, Colorado
  - Thornton, Colorado
  - Hamden, Connecticut
  - Jacksonville, Florida
  - Miami, Florida
  - Winter Park, Florida
  - Atlanta, Georgia
  - Decatur, Georgia
  - Macon, Georgia
  - Topeka, Kansas
  - Louisville, Kentucky
  - Baton Rouge, Louisiana
  - Chevy Chase, Maryland
  - Ann Arbor, Michigan
  - Troy, Michigan
  - Rochester, Minnesota
  - Cheektowaga, New York
  - New York, New York
  - Charlotte, North Carolina
  - Elkin, North Carolina
  - Portland, Oregon
  - Germantown, Tennessee
  - San Antonio, Texas
  - Tyler, Texas
  - Charlottesville, Virginia
  - Richmond, Virginia
  - Milwaukee, Wisconsin
- Adelaide, South Australia, Australia
- Leuven, Belgium
- Canada (2):
  - Edmonton, Alberta
  - Saskatoon, Saskatchewan
- Prague, Czechia
- Halle, Saint, Germany
- Szekszárd, Hungary
- Tel Aviv, Israel
- Kuala Lumpur, Malaysia
- Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/ For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Dulai PS, Feagan BG, Sands BE, Chen J, Lasch K, Lirio RA. Prognostic Value of Fecal Calprotectin to Inform Treat-to-Target Monitoring in Ulcerative Colitis. Clin Gastroenterol Hepatol. 2023 Feb;21(2):456-466.e7. doi: 10.1016/j.cgh.2022.07.027. Epub 2022 Aug 4. PMID 35934286
- [Derived] Wyant T, Yang L, Lirio RA, Rosario M. Vedolizumab Immunogenicity With Long-Term or Interrupted Treatment of Patients With Inflammatory Bowel Disease. J Clin Pharmacol. 2021 Sep;61(9):1174-1181. doi: 10.1002/jcph.1877. Epub 2021 Jul 14. PMID 33908636
- [Derived] Loftus EV Jr, Feagan BG, Panaccione R, Colombel JF, Sandborn WJ, Sands BE, Danese S, D'Haens G, Rubin DT, Shafran I, Parfionovas A, Rogers R, Lirio RA, Vermeire S. Long-term safety of vedolizumab for inflammatory bowel disease. Aliment Pharmacol Ther. 2020 Oct;52(8):1353-1365. doi: 10.1111/apt.16060. Epub 2020 Sep 2. PMID 32876349
- [Derived] Feagan BG, Schreiber S, Wolf DC, Axler JL, Kaviya A, James A, Curtis RI, Geransar P, Stallmach A, Ehehalt R, Bokemeyer B, Khalid JM, O'Byrne S. Sustained Clinical Remission With Vedolizumab in Patients With Moderate-to-Severe Ulcerative Colitis. Inflamm Bowel Dis. 2019 May 4;25(6):1028-1035. doi: 10.1093/ibd/izy323. PMID 30365009
- [Derived] Arijs I, De Hertogh G, Lemmens B, Van Lommel L, de Bruyn M, Vanhove W, Cleynen I, Machiels K, Ferrante M, Schuit F, Van Assche G, Rutgeerts P, Vermeire S. Effect of vedolizumab (anti-alpha4beta7-integrin) therapy on histological healing and mucosal gene expression in patients with UC. Gut. 2018 Jan;67(1):43-52. doi: 10.1136/gutjnl-2016-312293. Epub 2016 Oct 7. PMID 27802155
- [Derived] Colombel JF, Sands BE, Rutgeerts P, Sandborn W, Danese S, D'Haens G, Panaccione R, Loftus EV Jr, Sankoh S, Fox I, Parikh A, Milch C, Abhyankar B, Feagan BG. The safety of vedolizumab for ulcerative colitis and Crohn's disease. Gut. 2017 May;66(5):839-851. doi: 10.1136/gutjnl-2015-311079. Epub 2016 Feb 18. PMID 26893500

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in study at 298 sites in North America, Western/Northern Europe, Central Europe, Eastern Europe, Asia, Australia and Africa from 22 May 2009 to 31 October 2017.
Pre-assignment Details: Participants with a diagnosis of ulcerative colitis and Crohn's disease who participated in previous studies: C13004 (NCT00619489), C13006 (NCT00783718), C13007 (NCT00783692) and C13011 (NCT01224171) and DeNovo participants were enrolled into 1 treatment group, vedolizumab 300 mg, 30-minute intravenous (IV) infusion, every 4 weeks (Q4W).
Groups:
- Vedolizumab 300 mg (C13006): Vedolizumab 300 mg, 30-minute IV infusion, Q4W in this study. Treatment duration was up to approximately 430 weeks including treatment in the previous study. In study C13006: participants received either vedolizumab matching placebo or vedolizumab every Q4W or vedolizumab every 8 weeks (Q8W), IV infusion up to Week 52.
- Vedolizumab 300 mg (C13007): Vedolizumab 300 mg, 30-minute IV infusion, Q4W in this study. Treatment duration was up to approximately 429 weeks including treatment in the previous study. In study C13007: participants received either vedolizumab matching placebo or vedolizumab Q4W or vedolizumab Q8W, IV infusion up to Week 52.
- Vedolizumab 300 mg (C13011): Vedolizumab 300 mg, 30-minute IV infusion, Q4W in this study. Treatment duration was up to approximately 315 weeks including treatment in the previous study. In study C13011: participants received either vedolizumab matching placebo or vedolizumab 300 mg, IV infusion, at Weeks 0, 2 and 6.
- Vedolizumab 300 mg (C13004): Vedolizumab 300 mg, 30-minute IV infusion, Q4W in this study. Treatment duration was up to approximately 510 weeks including treatment in the previous study. In study C13004: participants received either vedolizumab 2 mg/kg or 6 mg/kg, IV infusion Q8W up to Week 78.
- Vedolizumab 300 mg (C13008 De Novo Participants): Vedolizumab 300 mg, 30-minute IV infusion, Q4W in this study. Treatment duration was up to approximately 260 weeks in participants with Crohn's disease (CD) or ulcerative colitis (UC) not treated in a previous study.
Period: Overall Study
Arm/Group | Vedolizumab 300 mg (C13006) | Vedolizumab 300 mg (C13007) | Vedolizumab 300 mg (C13011) | Vedolizumab 300 mg (C13004) | Vedolizumab 300 mg (C13008 De Novo Participants)
Started | 675 | 726 | 384 | 37 | 421
Completed | 237 | 246 | 115 | 23 | 145
Not Completed | 438 | 480 | 269 | 14 | 276
Not completed — Adverse Event | 94 | 119 | 65 | 5 | 69
Not completed — Protocol Violation(s) | 8 | 18 | 7 | 0 | 12
Not completed — Lack of Efficacy | 192 | 176 | 130 | 1 | 121
Not completed — Study Terminated by Sponsor | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 123 | 120 | 52 | 6 | 50
Not completed — Lost to Follow-up | 13 | 31 | 10 | 1 | 15
Not completed — Reason Not Specified | 8 | 16 | 4 | 1 | 9

BASELINE CHARACTERISTICS:
Population: Safety population was defined as all participants who received any amount of vedolizumab in this study.
Groups:
- Vedolizumab 300 mg (C13006): Vedolizumab 300 mg, 30-minute IV infusion, Q4W in this study. Treatment duration was up to approximately 430 weeks including treatment in the previous study. In study C13006: participants received either vedolizumab matching placebo or vedolizumab every Q4W or vedolizumab Q8W, IV infusion up to Week 52.
- Total: Total of all reporting groups
Arm/Group | Vedolizumab 300 mg (C13006) | Vedolizumab 300 mg (C13007) | Vedolizumab 300 mg (C13011) | Vedolizumab 300 mg (C13004) | Vedolizumab 300 mg (C13008 De Novo Participants) | Total
Number analyzed (Participants) | 675 | 726 | 384 | 37 | 421 | 2243
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.2 (13.27) | 37.3 (12.26) | 38.3 (12.87) | 43.9 (14.24) | 39.3 (14.23) | 39.1 (13.19)
Age, Customized [Count of Participants; unit: Participants]
  <65 | 646 | 710 | 376 | 35 | 400 | 2167
  >=65 | 29 | 16 | 8 | 2 | 21 | 76
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 280 | 384 | 216 | 20 | 215 | 1115
  Male | 395 | 342 | 168 | 17 | 206 | 1128
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 29 | 12 | 7 | 0 | 19 | 67
  Not Hispanic or Latino | 631 | 700 | 372 | 36 | 400 | 2139
  Unknown or Not Reported | 15 | 14 | 5 | 1 | 2 | 37
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 557 | 641 | 349 | 36 | 398 | 1981
  Black | 10 | 17 | 7 | 0 | 8 | 42
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 1 | 0 | 0 | 3
  Asian | 98 | 66 | 14 | 0 | 9 | 187
  American Indian or Alaskan Native | 2 | 0 | 0 | 1 | 0 | 3
  Other | 6 | 2 | 11 | 0 | 5 | 24
  Not Reported | 0 | 0 | 2 | 0 | 1 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  Australia | 41 | 30 | 8 | 0 | 21 | 100
  Hong Kong | 1 | 2 | 0 | 0 | 0 | 3
  India | 39 | 24 | 0 | 0 | 0 | 63
  Malaysia | 8 | 6 | 3 | 0 | 0 | 17
  New Zealand | 9 | 8 | 1 | 0 | 8 | 26
  Singapore | 1 | 1 | 0 | 0 | 0 | 2
  South Africa | 13 | 15 | 8 | 0 | 0 | 36
  Korea, Republic Of | 34 | 18 | 7 | 0 | 0 | 59
  Taiwan, Province Of China | 1 | 3 | 0 | 0 | 0 | 4
  Czech Republic | 34 | 67 | 36 | 0 | 69 | 206
  Greece | 5 | 0 | 0 | 0 | 0 | 5
  Hungary | 12 | 47 | 22 | 0 | 17 | 98
  Poland | 53 | 20 | 9 | 0 | 0 | 82
  Romania | 0 | 4 | 0 | 0 | 0 | 4
  Serbia | 0 | 2 | 0 | 0 | 0 | 2
  Slovakia | 0 | 14 | 17 | 0 | 0 | 31
  Bulgaria | 5 | 6 | 0 | 0 | 0 | 11
  Estonia | 9 | 5 | 0 | 0 | 0 | 14
  Israel | 2 | 12 | 21 | 0 | 21 | 56
  Latvia | 0 | 1 | 0 | 0 | 0 | 1
  Russia | 46 | 24 | 0 | 15 | 0 | 85
  Turkey | 6 | 3 | 0 | 0 | 0 | 9
  Ukraine | 0 | 9 | 0 | 0 | 0 | 9
  Canada | 73 | 98 | 75 | 22 | 87 | 355
  United States | 169 | 166 | 109 | 0 | 147 | 591
  Austria | 13 | 9 | 3 | 0 | 0 | 25
  Belgium | 48 | 48 | 33 | 0 | 46 | 175
  Denmark | 2 | 0 | 0 | 0 | 0 | 2
  France | 11 | 25 | 10 | 0 | 0 | 46
  Germany | 10 | 25 | 4 | 0 | 5 | 44
  Iceland | 3 | 3 | 0 | 0 | 0 | 6
  Ireland | 1 | 1 | 0 | 0 | 0 | 2
  Italy | 12 | 7 | 4 | 0 | 0 | 23
  Netherlands | 2 | 5 | 12 | 0 | 0 | 19
  Norway | 7 | 5 | 2 | 0 | 0 | 14
  Spain | 1 | 4 | 0 | 0 | 0 | 5
  Sweden | 0 | 5 | 0 | 0 | 0 | 5
  Switzerland | 2 | 4 | 0 | 0 | 0 | 6
  United Kingdom | 2 | 0 | 0 | 0 | 0 | 2
Body Weight [Mean (Standard Deviation); unit: kg] | 74.10 (17.934) | 71.70 (19.600) | 71.29 (18.951) | 77.66 (18.907) | 75.45 (18.814) | 73.15 (18.900)
BMI [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index = weight (kg)/[height (m)^2]. BMI was not calculated for de novo participants as height was not collected for these participants. BMI data was available for only 1822 participants. Population: BMI was not calculated for de novo participants due to no collection of height information.
  kg/m^2
    number analyzed (Participants) | 675 | 726 | 384 | 37 | 0 | 1822
    (all) | 25.39 (5.391) | 24.61 (6.039) | 24.56 (5.783) | 27.11 (6.523) |  | 24.94 (5.779)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With One or More Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An adverse event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (eg, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A treatment-emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs after receiving study drug. A serious adverse event (SAE) is any experience that suggests a significant hazard, contraindication, side effect or precaution that: results in death, is life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or is medically significant.
Time Frame: From first dose of study drug in this study through 16 weeks after the last dose of study drug (Up to approximately 8.5 years)
Population: The safety population was defined as all participants who participated in Studies C13004, C13006, C13007, and C13011 and received any amount of vedolizumab in Study C13008. De novo participants who received any amount of vedolizumab in Study C13008 were also included in the safety population.
Measure: Number; unit: percentage of participants
Groups:
- Vedolizumab 300 mg (UC): Vedolizumab 300 mg, 30-minute IV infusion, Q4W, up to approximately 260 weeks. Includes De Novo participants and participants previously enrolled in studies C13004 and C13006 with a diagnosis of Ulcerative colitis (UC).
- Vedolizumab 300 mg (CD): Vedolizumab 300 mg, 30-minute IV infusion, Q4W, up to approximately 260 weeks. Includes De Novo participants and participants previously enrolled in studies C13004, C13007 and C13011 with a diagnosis of Crohn's disease.
Arm/Group | Vedolizumab 300 mg (UC) | Vedolizumab 300 mg (CD)
Number analyzed (Participants) | 894 | 1349
percentage of participants
  TEAEs | 93 | 96
  SAEs | 31 | 41

2. Primary Outcome: Number of Participants With Markedly Abnormal Safety Laboratory Findings
Description: A laboratory value was considered a marked abnormality if it met the predefined criteria or parameters and the on-treatment value was more extreme than the Baseline value for the following parameters: hemoglobin <= 70 g/L, absolute lymphocyte count <0.5 X 10^9/L, leukocytes <2.0 X 10^9/L (absolute value), platelets <75.0 X 10^9/L, absolute neutrophil Count <1.0 X 10^9/L, prothrombin time >1.25 x upper limit of normal (ULN), alanine aminotransferase (ALT) >3.0 x ULN, aspartate aminotransferase (AST) >3.0 x ULN, bilirubin >2.0 x ULN, amylase >2.0 x ULN, lipase >2.0 x ULN.
Time Frame: From first dose of study drug in this study through 16 weeks after the last dose of study drug (Up to 8.5 years)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Vedolizumab 300 mg (UC) | Vedolizumab 300 mg (CD)
Number analyzed (Participants) | 894 | 1349
participants
  Hemoglobin <= 70 g/L | 16 | 11
  Absolute Lymphocyte Count <0.5 X 10^9/L | 28 | 56
  Leukocytes <2.0 X 10^9/L (Absolute Value) | 1 | 3
  Platelets <75.0 X 10^9/L | 2 | 5
  Absolute Neutrophil Count <1.0 X 10^9/L | 9 | 9
  Prothrombin Time >1.25 x ULN | 42 | 37
  ALT >3.0 x ULN | 30 | 47
  AST >3.0 x ULN | 35 | 34
  Bilirubin >2.0 x ULN | 12 | 14
  Amylase >2.0 x ULN | 16 | 36
  Lipase >2.0 x ULN | 27 | 41

3. Primary Outcome: Percentage of Participants With at Least One Clinically Significant Mean Change Over Time in Vital Sign Measurements
Description: Vital signs (heart rate, respiratory rate, systolic and diastolic blood pressure, and temperature) measurements were collected throughout the study. Any clinically significant mean change in vital signs over time as assessed by the investigator was reported as a TEAE.
Time Frame: From first dose of study drug in this study through 16 weeks after the last dose of study drug (Up to 8.5 years)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Vedolizumab 300 mg (UC) | Vedolizumab 300 mg (CD)
Number analyzed (Participants) | 894 | 1349
percentage of participants | 0 | 0

4. Primary Outcome: Number of Participants With at Least One Clinically Significant Electrocardiogram (ECG) Findings
Description: A standard 12-lead ECG was performed. Any ECGs assessed by the investigator to be clinically significant were reported as TEAEs.
Time Frame: From first dose of study drug in this study through 16 weeks after the last dose of study drug (Up to 8.5 years)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Vedolizumab 300 mg (UC) | Vedolizumab 300 mg (CD)
Number analyzed (Participants) | 894 | 1349
participants | 7 | 7

5. Primary Outcome: Time to Major Inflammatory Bowel Disease (IBD) - Related Events
Description: IBD-related events included hospitalizations, surgeries, or procedures due to ulcerative colitis and Crohn's disease.
Time Frame: Baseline (Prior to first dose of study drug in C13008) up to end of study (approximately up to 8.5 years)
Population: Efficacy population included participants who received at least one dose of vedolizumab and had at least one postbaseline disease activity measurement.
Measure: Median (95% Confidence Interval); unit: weeks
Groups:
- Vedolizumab 300 mg: Vedolizumab 300 mg, 30-minute IV infusion, Q4W, up to approximately 260 weeks.
Arm/Group | Vedolizumab 300 mg
Number analyzed (Participants) | 2142
weeks
  IBD-related events, UC: number analyzed (Participants) | 845
  IBD-related events, UC | NA [NA to NA] — Median was not estimable due to the low number of participants with events.
  IBD-related events, CD: number analyzed (Participants) | 1297
  IBD-related events, CD | NA [NA to NA] — Median was not estimable due to the low number of participants with events.

6. Primary Outcome: Change From Baseline in the Inflammatory Bowel Disease Questionnaire (IBDQ) Scores at Week 28
Description: The IBDQ is an instrument used to assess quality of life in adult participants with inflammatory bowel disease (IBD). It includes 32 questions on 4 domains of Health-Related Quality-of-Life (HRQOL): Bowel Systems (10 items), Emotional Function (12 items), Social Function (5 items), and Systemic Function (5 items). Participants are asked to recall symptoms and quality of life from the last 2 weeks and rate each item on a 7-point Likert scale (1=worst to 7=best). A total IBDQ score is calculated by summing the scores from each domain; the total IBDQ score ranges from 32 to 224, with lower scores reflecting worse HRQOL. A positive change from Baseline indicates improvement.
Time Frame: Baseline (prior to first dose of study drug in C13008; for rollover participants this was the last assessment from the previous study) and Week 28
Population: Intent to treat (ITT) population from studies C13006, C13007, C13011 and de novo participants who received vedolizumab in study C13008. Data is provided for participants who were completers in previous studies and de novo participants for whom data was collected at both Baseline and Week 28. Not applicable for Vedolizumab 300 mg (C13004) arm group.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Vedolizumab 300 mg (C13006 Placebo): Vedolizumab 300 mg, 30-minute IV infusion, Q4W in this study. Treatment duration was up to approximately 430 weeks including treatment in the previous study. In study C13006: vedolizumab matching placebo, IV infusion at Weeks 0 and 2 (Days 1 and 15). Participants continued to receive placebo during the Maintenance Phase, regardless of treatment response during Induction phase up to Week 50.
- Vedolizumab 300 mg (C13006 Vedolizumab Q8W): Vedolizumab 300 mg, 30-minute IV infusion, Q4W in this study. Treatment duration was up to approximately 430 weeks including treatment in the previous study. In study C13006: vedolizumab 300 mg, intravenous infusion at Weeks 0 and 2 (Days 1 and 15) in Induction Phase.
  In the Maintenance Phase, participants who demonstrated a clinical response at Week 6 according to protocol-specified criteria received vedolizumab, IV infusion, Q8W up to Week 50.
- Vedolizumab 300 mg (C13006 Vedolizumab Q4W): Vedolizumab 300 mg, 30-minute IV infusion, Q4W in this study. Treatment duration was up to approximately 430 weeks including treatment in the previous study. In study C13006: vedolizumab 300 mg, intravenous infusion at Week 0 and Week 2 (Days 1 and 15) in Induction Phase. In the Maintenance Phase, participants who demonstrated a clinical response at Week 6 according to protocol-specified criteria received vedolizumab, IV infusion, Q4W up to Week 50.
- Vedolizumab 300 mg (C13007 Placebo): Vedolizumab 300 mg, 30-minute IV infusion, Q4W in this study. Treatment duration was up to approximately 429 weeks including treatment in the previous study. In study C13007: vedolizumab matching placebo, intravenous infusion at Weeks 0 and 2 (Days 1 and 15). Participants continued to receive placebo during the Maintenance Phase, regardless of treatment response during Induction up to Week 52.
- Vedolizumab 300 mg (C13007 Vedolizumab Q8W): Vedolizumab 300 mg, 30-minute IV infusion, Q4W in this study. Treatment duration was up to approximately 429 weeks including treatment in the previous study. In study C13007: vedolizumab 300 mg, IV infusion at Weeks 0 and 2 (Days 1 and 15) in Induction Phase. In the Maintenance Phase, participants who demonstrated a clinical response at Week 6 according to protocol-specified criteria received vedolizumab, IV infusion, Q8W up to Week 52.
- Vedolizumab 300 mg (C13007 Vedolizumab Q4W): Vedolizumab 300 mg, 30-minute IV infusion, Q4W in this study. Treatment duration was up to approximately 429 weeks including treatment in the previous study. In study C13007: vedolizumab 300 mg, intravenous infusion at Weeks 0 and 2 (Days 1 and 15) in Induction Phase. In the Maintenance Phase, participants who demonstrated a clinical response at Week 6 according to protocol-specified criteria received vedolizumab, IV infusion, Q4W up to Week 52.
- Vedolizumab 300 mg (C13011 Placebo): Vedolizumab 300 mg, 30-minute IV infusion, Q4W in this study. Treatment duration was up to approximately 315 weeks including treatment in the previous study. In study C13011: vedolizumab matching placebo, IV infusion at Weeks 0, 2 and 6.
- Vedolizumab 300 mg (C13011 Vedolizumab): Vedolizumab 300 mg, 30-minute IV infusion, Q4W in this study. Treatment duration was up to approximately up to 315 weeks including treatment in the previous study. In study C13011: vedolizumab 300 mg, IV infusion, at Weeks 0, 2 and 6.
- Vedolizumab 300 mg (C13008 De Novo Participants - UC): Vedolizumab 300 mg, 30-minute IV infusion, Q4W, up to approximately 260 weeks in participants with ulcerative colitis not treated in previous study.
- Vedolizumab 300 mg (C13008 De Novo Participants - CD): Vedolizumab 300 mg, 30-minute IV infusion, Q4W, starting at Week 0, up to approximately 260 weeks in participants with Crohn's disease not treated in a previous study.
Arm/Group | Vedolizumab 300 mg (C13006 Placebo) | Vedolizumab 300 mg (C13006 Vedolizumab Q8W) | Vedolizumab 300 mg (C13006 Vedolizumab Q4W) | Vedolizumab 300 mg (C13007 Placebo) | Vedolizumab 300 mg (C13007 Vedolizumab Q8W) | Vedolizumab 300 mg (C13007 Vedolizumab Q4W) | Vedolizumab 300 mg (C13011 Placebo) | Vedolizumab 300 mg (C13011 Vedolizumab) | Vedolizumab 300 mg (C13008 De Novo Participants - UC) | Vedolizumab 300 mg (C13008 De Novo Participants - CD)
Number analyzed (Participants) | 38 | 67 | 76 | 52 | 62 | 71 | 127 | 134 | 150 | 161
score on a scale
  Baseline | 125.34 (34.895) | 129.12 (34.289) | 124.37 (31.632) | 122.33 (31.114) | 127.56 (33.718) | 127.11 (30.537) | 123.88 (31.620) | 124.35 (33.310) | 131.44 (27.715) | 132.14 (32.245)
  Change at Week 28 | 60.00 (41.165) | 62.71 (34.600) | 62.53 (35.072) | 57.17 (38.851) | 57.52 (42.561) | 51.48 (34.576) | 41.71 (36.508) | 40.49 (39.733) | 42.90 (32.581) | 30.84 (34.614)

7. Primary Outcome: Change From Baseline in the Inflammatory Bowel Disease Questionnaire (IBDQ) Scores at Week 52
Description: as for outcome 6
Time Frame: Baseline (prior to first dose of study drug in C13008; for rollover participants this was the last assessment from the previous study) and Week 52
Population: The ITT population from studies C13006, C13007, C13011 and de novo participants who received vedolizumab in study C13008. Data is provided for participants who were completers in previous studies and de novo participants for whom data was collected at both Baseline and Week 52. Not applicable for Vedolizumab 300 mg (C13004) arm group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vedolizumab 300 mg (C13006 Placebo) | Vedolizumab 300 mg (C13006 Vedolizumab Q8W) | Vedolizumab 300 mg (C13006 Vedolizumab Q4W) | Vedolizumab 300 mg (C13007 Placebo) | Vedolizumab 300 mg (C13007 Vedolizumab Q8W) | Vedolizumab 300 mg (C13007 Vedolizumab Q4W) | Vedolizumab 300 mg (C13011 Placebo) | Vedolizumab 300 mg (C13011 Vedolizumab) | Vedolizumab 300 mg (C13008 De Novo Participants - UC) | Vedolizumab 300 mg (C13008 De Novo Participants - CD)
Number analyzed (Participants) | 32 | 65 | 70 | 49 | 56 | 63 | 107 | 117 | 132 | 134
score on a scale
  Baseline | 123.53 (36.160) | 131.17 (33.675) | 125.03 (32.560) | 120.29 (30.894) | 129.46 (34.799) | 128.69 (30.461) | 125.30 (30.075) | 125.31 (34.140) | 130.63 (28.446) | 132.71 (33.108)
  Change at Week 52 | 66.84 (41.733) | 59.89 (33.170) | 61.06 (37.386) | 59.31 (34.837) | 58.87 (40.707) | 52.30 (29.385) | 44.31 (37.923) | 47.38 (37.687) | 47.07 (30.463) | 37.33 (40.232)

8. Primary Outcome: Change From Baseline in the Inflammatory Bowel Disease Questionnaire (IBDQ) Scores at Week 76
Description: as for outcome 6
Time Frame: Baseline (prior to first dose of study drug in C13008; for rollover participants this was the last assessment from the previous study) and Week 76
Population: The ITT population from studies C13006, C13007, C13011 and de novo participants who received vedolizumab in study C13008. Data is provided for participants who were completers in previous studies and de novo participants for whom data was collected at both Baseline and Week 76. Not applicable for Vedolizumab 300 mg (C13004) arm group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vedolizumab 300 mg (C13006 Placebo) | Vedolizumab 300 mg (C13006 Vedolizumab Q8W) | Vedolizumab 300 mg (C13006 Vedolizumab Q4W) | Vedolizumab 300 mg (C13007 Placebo) | Vedolizumab 300 mg (C13007 Vedolizumab Q8W) | Vedolizumab 300 mg (C13007 Vedolizumab Q4W) | Vedolizumab 300 mg (C13011 Placebo) | Vedolizumab 300 mg (C13011 Vedolizumab) | Vedolizumab 300 mg (C13008 De Novo Participants - UC) | Vedolizumab 300 mg (C13008 De Novo Participants - CD)
Number analyzed (Participants) | 29 | 63 | 63 | 45 | 55 | 58 | 91 | 106 | 118 | 113
score on a scale
  Baseline | 123.66 (36.115) | 131.31 (33.726) | 123.87 (31.752) | 120.00 (29.667) | 128.47 (34.724) | 129.06 (31.694) | 124.89 (31.629) | 125.89 (34.478) | 130.75 (28.587) | 132.46 (33.245)
  Change at Week 76 | 65.53 (40.584) | 59.88 (35.290) | 64.27 (32.443) | 59.91 (34.449) | 55.05 (47.181) | 52.85 (36.486) | 47.43 (35.811) | 46.32 (36.397) | 50.59 (30.794) | 40.14 (39.305)

9. Primary Outcome: Change From Baseline in the Inflammatory Bowel Disease Questionnaire (IBDQ) Scores at Week 100
Description: as for outcome 6
Time Frame: Baseline (prior to first dose of study drug in C13008; for rollover participants this was the last assessment from the previous study) and Week 100
Population: The ITT population from studies C13006, C13007, C13011 and de novo participants who received vedolizumab in study C13008. Data is provided for participants who were completers in previous studies and de novo participants for whom data was collected at both Baseline and Week 100. Not applicable for Vedolizumab 300 mg (C13004) arm group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vedolizumab 300 mg (C13006 Placebo) | Vedolizumab 300 mg (C13006 Vedolizumab Q8W) | Vedolizumab 300 mg (C13006 Vedolizumab Q4W) | Vedolizumab 300 mg (C13007 Placebo) | Vedolizumab 300 mg (C13007 Vedolizumab Q8W) | Vedolizumab 300 mg (C13007 Vedolizumab Q4W) | Vedolizumab 300 mg (C13011 Placebo) | Vedolizumab 300 mg (C13011 Vedolizumab) | Vedolizumab 300 mg (C13008 De Novo Participants - UC) | Vedolizumab 300 mg (C13008 De Novo Participants - CD)
Number analyzed (Participants) | 27 | 58 | 58 | 45 | 49 | 55 | 84 | 96 | 112 | 104
score on a scale
  Baseline | 124.70 (37.614) | 130.90 (34.361) | 124.52 (30.033) | 120.89 (29.745) | 129.53 (35.261) | 128.25 (32.333) | 123.50 (29.662) | 128.35 (33.793) | 132.41 (28.538) | 132.48 (32.305)
  Change at Week 100 | 61.83 (41.505) | 62.46 (32.502) | 62.83 (34.475) | 57.04 (38.448) | 58.53 (45.644) | 53.40 (32.651) | 49.89 (36.806) | 46.95 (34.691) | 52.50 (32.267) | 38.52 (36.982)

10. Primary Outcome: Change From Baseline in the Inflammatory Bowel Disease Questionnaire (IBDQ) Scores at Week 124
Description: as for outcome 6
Time Frame: Baseline (prior to first dose of study drug in C13008; for rollover participants this was the last assessment from the previous study) and Week 124
Population: The ITT population from studies C13006, C13007, C13011 and de novo participants who received vedolizumab in study C13008. Data is provided for participants who were completers in previous studies and de novo participants for whom data was collected at both Baseline and Week 124. Not applicable for Vedolizumab 300 mg (C13004) arm group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vedolizumab 300 mg (C13006 Placebo) | Vedolizumab 300 mg (C13006 Vedolizumab Q8W) | Vedolizumab 300 mg (C13006 Vedolizumab Q4W) | Vedolizumab 300 mg (C13007 Placebo) | Vedolizumab 300 mg (C13007 Vedolizumab Q8W) | Vedolizumab 300 mg (C13007 Vedolizumab Q4W) | Vedolizumab 300 mg (C13011 Placebo) | Vedolizumab 300 mg (C13011 Vedolizumab) | Vedolizumab 300 mg (C13008 De Novo Participants - UC) | Vedolizumab 300 mg (C13008 De Novo Participants - CD)
Number analyzed (Participants) | 27 | 58 | 54 | 43 | 47 | 48 | 80 | 82 | 95 | 97
score on a scale
  Baseline | 127.33 (36.470) | 130.83 (34.399) | 123.65 (30.180) | 119.77 (29.963) | 132.36 (34.573) | 130.01 (33.454) | 122.91 (29.869) | 129.08 (33.576) | 132.75 (28.131) | 131.56 (31.567)
  Change at Week 124 | 63.94 (44.480) | 60.94 (37.769) | 63.71 (34.542) | 61.91 (36.288) | 53.91 (44.023) | 53.74 (34.514) | 46.62 (38.435) | 47.60 (40.634) | 54.47 (29.636) | 40.35 (41.543)

11. Primary Outcome: Change From Baseline in the Inflammatory Bowel Disease Questionnaire (IBDQ) Scores at Week 148
Description: as for outcome 6
Time Frame: Baseline (prior to first dose of study drug in C13008; for rollover participants this was the last assessment from the previous study) and Week 148
Population: The ITT population from studies C13006, C13007, C13011 and de novo participants who received vedolizumab in study C13008. Data is provided for participants who were completers in previous studies and de novo participants for whom data was collected at both Baseline and Week 148. Not applicable for Vedolizumab 300 mg (C13004) arm group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vedolizumab 300 mg (C13006 Placebo) | Vedolizumab 300 mg (C13006 Vedolizumab Q8W) | Vedolizumab 300 mg (C13006 Vedolizumab Q4W) | Vedolizumab 300 mg (C13007 Placebo) | Vedolizumab 300 mg (C13007 Vedolizumab Q8W) | Vedolizumab 300 mg (C13007 Vedolizumab Q4W) | Vedolizumab 300 mg (C13011 Placebo) | Vedolizumab 300 mg (C13011 Vedolizumab) | Vedolizumab 300 mg (C13008 De Novo Participants - UC) | Vedolizumab 300 mg (C13008 De Novo Participants - CD)
Number analyzed (Participants) | 27 | 54 | 53 | 41 | 43 | 46 | 76 | 83 | 93 | 92
score on a scale
  Baseline | 127.33 (36.470) | 131.95 (34.649) | 123.02 (29.685) | 119.07 (30.344) | 132.23 (35.877) | 130.25 (34.108) | 122.01 (28.967) | 128.66 (34.624) | 133.36 (28.616) | 132.38 (32.172)
  Change at Week 148 | 60.66 (41.786) | 62.72 (33.786) | 65.81 (33.232) | 60.41 (36.074) | 54.53 (48.036) | 56.08 (32.954) | 52.30 (39.123) | 49.40 (36.880) | 54.50 (32.874) | 42.13 (40.030)

12. Primary Outcome: Change From Baseline in the Inflammatory Bowel Disease Questionnaire (IBDQ) Scores at Week 172
Description: as for outcome 6
Time Frame: Baseline (prior to first dose of study drug in C13008; for rollover participants this was the last assessment from the previous study) and Week 172
Population: The ITT population from studies C13006, C13007, C13011 and de novo participants who received vedolizumab in study C13008. Data is provided for participants who were completers in previous studies and de novo participants for whom data was collected at both Baseline and Week 172. Not applicable for Vedolizumab 300 mg (C13004) arm group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vedolizumab 300 mg (C13006 Placebo) | Vedolizumab 300 mg (C13006 Vedolizumab Q8W) | Vedolizumab 300 mg (C13006 Vedolizumab Q4W) | Vedolizumab 300 mg (C13007 Placebo) | Vedolizumab 300 mg (C13007 Vedolizumab Q8W) | Vedolizumab 300 mg (C13007 Vedolizumab Q4W) | Vedolizumab 300 mg (C13011 Placebo) | Vedolizumab 300 mg (C13011 Vedolizumab) | Vedolizumab 300 mg (C13008 De Novo Participants - UC) | Vedolizumab 300 mg (C13008 De Novo Participants - CD)
Number analyzed (Participants) | 24 | 53 | 49 | 37 | 43 | 43 | 71 | 76 | 89 | 80
score on a scale
  Baseline | 130.25 (36.650) | 132.93 (34.216) | 123.47 (30.141) | 120.49 (30.221) | 131.60 (36.013) | 132.31 (33.860) | 120.70 (27.535) | 127.42 (34.779) | 133.34 (28.981) | 131.69 (32.229)
  Change at Week 172 | 58.67 (42.513) | 62.20 (33.187) | 62.16 (33.969) | 65.43 (35.350) | 54.91 (40.758) | 53.92 (33.132) | 51.55 (40.714) | 47.97 (35.121) | 56.02 (33.863) | 41.18 (40.805)

13. Primary Outcome: Change From Baseline in the Inflammatory Bowel Disease Questionnaire (IBDQ) Scores at Week 196
Description: as for outcome 6
Time Frame: Baseline (prior to first dose of study drug in C13008; for rollover participants this was the last assessment from the previous study) and Week 196
Population: The ITT population from studies C13006, C13007, C13011 and de novo participants who received vedolizumab in study C13008. Data is provided for participants who were completers in previous studies and de novo participants for whom data was collected at both Baseline and Week 196. Not applicable for Vedolizumab 300 mg (C13004) arm group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vedolizumab 300 mg (C13006 Placebo) | Vedolizumab 300 mg (C13006 Vedolizumab Q8W) | Vedolizumab 300 mg (C13006 Vedolizumab Q4W) | Vedolizumab 300 mg (C13007 Placebo) | Vedolizumab 300 mg (C13007 Vedolizumab Q8W) | Vedolizumab 300 mg (C13007 Vedolizumab Q4W) | Vedolizumab 300 mg (C13011 Placebo) | Vedolizumab 300 mg (C13011 Vedolizumab) | Vedolizumab 300 mg (C13008 De Novo Participants - UC) | Vedolizumab 300 mg (C13008 De Novo Participants - CD)
Number analyzed (Participants) | 27 | 50 | 46 | 37 | 41 | 41 | 66 | 71 | 62 | 51
score on a scale
  Baseline | 127.33 (36.470) | 135.33 (33.596) | 122.00 (30.129) | 119.35 (31.651) | 130.39 (36.410) | 132.16 (34.217) | 121.15 (28.703) | 126.44 (34.826) | 136.55 (27.551) | 137.27 (30.844)
  Change at Week 196 | 63.19 (38.061) | 59.13 (33.318) | 68.89 (34.578) | 64.81 (36.563) | 58.90 (46.107) | 55.67 (32.453) | 52.22 (42.363) | 49.41 (35.662) | 49.05 (30.390) | 36.35 (41.424)

14. Primary Outcome: Change From Baseline in the Inflammatory Bowel Disease Questionnaire (IBDQ) Scores at Week 248
Description: as for outcome 6
Time Frame: Baseline (prior to first dose of study drug in C13008; for rollover participants this was the last assessment from the previous study) and Week 248
Population: The ITT population from studies C13006, C13007, C13011 and de novo participants who received vedolizumab in study C13008. Data is provided for participants who were completers in previous studies and de novo participants for whom data was collected at both Baseline and Week 248. Not applicable for Vedolizumab 300 mg (C13004) arm group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vedolizumab 300 mg (C13006 Placebo) | Vedolizumab 300 mg (C13006 Vedolizumab Q8W) | Vedolizumab 300 mg (C13006 Vedolizumab Q4W) | Vedolizumab 300 mg (C13007 Placebo) | Vedolizumab 300 mg (C13007 Vedolizumab Q8W) | Vedolizumab 300 mg (C13007 Vedolizumab Q4W) | Vedolizumab 300 mg (C13011 Placebo) | Vedolizumab 300 mg (C13011 Vedolizumab) | Vedolizumab 300 mg (C13008 De Novo Participants - UC) | Vedolizumab 300 mg (C13008 De Novo Participants - CD)
Number analyzed (Participants) | 21 | 38 | 36 | 32 | 32 | 31 | 38 | 45 | 3 | 4
score on a scale
  Baseline | 116.05 (31.747) | 133.61 (32.538) | 120.28 (30.875) | 116.63 (32.888) | 131.81 (35.906) | 129.37 (31.455) | 122.00 (27.231) | 125.93 (35.080) | 127.00 (63.930) | 128.00 (35.749)
  Change at Week 248 | 76.21 (38.693) | 57.52 (31.841) | 69.56 (38.680) | 65.72 (34.776) | 54.97 (41.658) | 58.76 (35.250) | 51.39 (45.950) | 53.04 (38.830) | 73.00 (48.446) | 72.00 (32.156)

15. Primary Outcome: Change From Baseline in the Inflammatory Bowel Disease Questionnaire (IBDQ) Scores at Week 300
Description: as for outcome 6
Time Frame: Baseline (prior to first dose of study drug in C13008; for rollover participants this was the last assessment from the previous study) and Week 300
Population: ITT population from studies C13006, C13007 and C13011 who received vedolizumab in study C13008. Data is provided for participants who were completers in previous studies with data available at both Baseline and Week 300. Not applicable (NA) for Vedolizumab 300 mg (C13004) arm group. Data is not available for de novo participants at this time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vedolizumab 300 mg (C13006 Placebo) | Vedolizumab 300 mg (C13006 Vedolizumab Q8W) | Vedolizumab 300 mg (C13006 Vedolizumab Q4W) | Vedolizumab 300 mg (C13007 Placebo) | Vedolizumab 300 mg (C13007 Vedolizumab Q8W) | Vedolizumab 300 mg (C13007 Vedolizumab Q4W) | Vedolizumab 300 mg (C13011 Placebo) | Vedolizumab 300 mg (C13011 Vedolizumab)
Number analyzed (Participants) | 7 | 14 | 13 | 9 | 8 | 16 | 4 | 2
score on a scale
  Baseline | 100.71 (21.831) | 137.50 (30.478) | 120.38 (24.401) | 119.67 (33.463) | 134.88 (36.957) | 121.38 (30.133) | 120.25 (19.085) | 162.50 (47.376)
  Change at Week 300 | 94.29 (38.612) | 55.43 (41.694) | 67.54 (27.823) | 69.00 (41.192) | 53.00 (41.542) | 72.00 (35.219) | 73.50 (12.342) | 2.00 (5.657)

16. Primary Outcome: Change From Baseline in the Inflammatory Bowel Disease Questionnaire (IBDQ) Scores at Week 352
Description: as for outcome 6
Time Frame: Baseline (prior to first dose of study drug in C13008; for rollover participants this was the last assessment from the previous study) and Week 352
Population: ITT population from studies C13006 and C13007 who received vedolizumab in study C13008. Data is provided for completers in previous studies with data available at both Baseline and Week 352. NA for Vedolizumab 300 mg (C13004) arm group. Data is not available for C13011 Placebo and Vedolizumab arm groups and de novo participants at this time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vedolizumab 300 mg (C13006 Placebo) | Vedolizumab 300 mg (C13006 Vedolizumab Q8W) | Vedolizumab 300 mg (C13006 Vedolizumab Q4W) | Vedolizumab 300 mg (C13007 Placebo) | Vedolizumab 300 mg (C13007 Vedolizumab Q8W) | Vedolizumab 300 mg (C13007 Vedolizumab Q4W)
Number analyzed (Participants) | 1 | 1 | 3 | 1 | 2 | 1
score on a scale
  Baseline | 89.00 (NA) — Standard deviation (SD) was not calculated for 1 participant. | 120.00 (NA) — SD was not calculated for 1 participant. | 118.00 (32.047) | 70.00 (NA) — SD was not calculated for 1 participant. | 137.00 (28.284) | 126.00 (NA) — SD was not calculated for 1 participant.
  Change at Week 352 | 123.00 (NA) — SD was not calculated for 1 participant. | 86.00 (NA) — SD was not calculated for 1 participant. | 66.00 (33.181) | 131.00 (NA) — SD was not calculated for 1 participant. | 37.50 (28.991) | 84.00 (NA) — SD was not calculated for 1 participant.

17. Primary Outcome: Change From Baseline in Short Form-36 (SF-36) Physical Component Scores at Week 28
Description: The Short Form-36 (SF-36) is a questionnaire that evaluates a person's HRQOL. SF-36 includes 36 questions related to 8 health dimensions: physical functioning, role-physical (role limitations due to physical health problems), bodily pain, general health, vitality (energy/fatigue), social functioning, role-emotional (role limitations due to emotional problems), and mental health. Based on these 4 scales (physical functioning, role-physical, bodily pain, general health), the physical component summary (PCS) score is generated which ranges between 0 and 100, with higher scores indicating a better quality of life. A positive change from Baseline indicates improvement.
Time Frame: as for outcome 6
Population: The ITT population from studies C13006, C13007, C13011 and de novo participants who received vedolizumab in study C13008. Data is provided for participants who were completers in previous studies and de novo participants for whom data was collected at both Baseline and Week 28. Not applicable for Vedolizumab 300 mg (C13004) arm group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vedolizumab 300 mg (C13006 Placebo) | Vedolizumab 300 mg (C13006 Vedolizumab Q8W) | Vedolizumab 300 mg (C13006 Vedolizumab Q4W) | Vedolizumab 300 mg (C13007 Placebo) | Vedolizumab 300 mg (C13007 Vedolizumab Q8W) | Vedolizumab 300 mg (C13007 Vedolizumab Q4W) | Vedolizumab 300 mg (C13011 Placebo) | Vedolizumab 300 mg (C13011 Vedolizumab) | Vedolizumab 300 mg (C13008 De Novo Participants - UC) | Vedolizumab 300 mg (C13008 De Novo Participants - CD)
Number analyzed (Participants) | 38 | 67 | 76 | 52 | 62 | 71 | 127 | 136 | 151 | 162
score on a scale
  Baseline | 39.57 (8.599) | 41.15 (8.313) | 40.05 (7.634) | 37.05 (7.522) | 37.87 (8.113) | 39.09 (7.771) | 37.92 (8.355) | 36.81 (8.274) | 40.06 (8.631) | 39.20 (7.306)
  Change at Week 28 | 10.20 (8.792) | 8.22 (9.015) | 8.89 (7.110) | 9.85 (8.789) | 12.46 (8.900) | 9.60 (7.620) | 6.48 (8.514) | 7.74 (9.310) | 7.07 (8.752) | 5.67 (7.695)

18. Primary Outcome: Change From Baseline in Short Form-36 (SF-36) Mental Component Scores at Week 28
Description: The Short Form-36 (SF-36) is a questionnaire that evaluates a person's HRQOL. SF-36 includes 36 questions related to 8 health dimensions: physical functioning, role-physical (role limitations due to physical health problems), bodily pain, general health, vitality (energy/fatigue), social functioning, role-emotional (role limitations due to emotional problems), and mental health. Based on these 4 scales (vitality, social functioning, role-emotional, and mental health), the mental component summary (MCS) score is generated which ranges between 0 and 100, with higher scores indicating a better quality of life. A positive change from Baseline indicates improvement.
Time Frame: as for outcome 6
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vedolizumab 300 mg (C13006 Placebo) | Vedolizumab 300 mg (C13006 Vedolizumab Q8W) | Vedolizumab 300 mg (C13006 Vedolizumab Q4W) | Vedolizumab 300 mg (C13007 Placebo) | Vedolizumab 300 mg (C13007 Vedolizumab Q8W) | Vedolizumab 300 mg (C13007 Vedolizumab Q4W) | Vedolizumab 300 mg (C13011 Placebo) | Vedolizumab 300 mg (C13011 Vedolizumab) | Vedolizumab 300 mg (C13008 De Novo Participants - UC) | Vedolizumab 300 mg (C13008 De Novo Participants - CD)
Number analyzed (Participants) | 38 | 67 | 76 | 52 | 62 | 71 | 127 | 136 | 151 | 162
score on a scale
  Baseline | 39.98 (11.349) | 40.70 (11.226) | 38.28 (11.039) | 35.49 (11.139) | 38.53 (10.631) | 37.70 (12.423) | 36.60 (11.545) | 38.04 (12.567) | 40.87 (11.385) | 39.29 (11.535)
  Change at Week 28 | 8.36 (13.096) | 11.10 (11.098) | 11.52 (12.464) | 13.35 (11.857) | 10.88 (12.396) | 10.94 (12.386) | 7.48 (12.061) | 6.34 (13.161) | 6.48 (10.809) | 3.72 (12.377)

19. Primary Outcome: Change From Baseline in Short Form-36 (SF-36) Physical Component Score at Week 52
Description: as for outcome 17
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vedolizumab 300 mg (C13006 Placebo) | Vedolizumab 300 mg (C13006 Vedolizumab Q8W) | Vedolizumab 300 mg (C13006 Vedolizumab Q4W) | Vedolizumab 300 mg (C13007 Placebo) | Vedolizumab 300 mg (C13007 Vedolizumab Q8W) | Vedolizumab 300 mg (C13007 Vedolizumab Q4W) | Vedolizumab 300 mg (C13011 Placebo) | Vedolizumab 300 mg (C13011 Vedolizumab) | Vedolizumab 300 mg (C13008 De Novo Participants - UC) | Vedolizumab 300 mg (C13008 De Novo Participants - CD)
Number analyzed (Participants) | 32 | 64 | 69 | 49 | 56 | 63 | 107 | 118 | 133 | 135
score on a scale
  Baseline | 39.94 (8.930) | 41.72 (8.314) | 40.12 (7.694) | 36.75 (7.510) | 37.82 (8.301) | 39.23 (7.807) | 37.87 (7.992) | 37.40 (8.171) | 40.51 (8.454) | 39.27 (7.469)
  Change at Week 52 | 9.55 (10.155) | 8.57 (7.889) | 9.77 (6.766) | 9.43 (9.088) | 12.97 (9.147) | 9.98 (7.824) | 7.48 (8.800) | 8.97 (8.743) | 8.37 (8.401) | 6.72 (7.842)

20. Primary Outcome: Change From Baseline in Short Form-36 (SF-36) Mental Component Score at Week 52
Description: as for outcome 18
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vedolizumab 300 mg (C13006 Placebo) | Vedolizumab 300 mg (C13006 Vedolizumab Q8W) | Vedolizumab 300 mg (C13006 Vedolizumab Q4W) | Vedolizumab 300 mg (C13007 Placebo) | Vedolizumab 300 mg (C13007 Vedolizumab Q8W) | Vedolizumab 300 mg (C13007 Vedolizumab Q4W) | Vedolizumab 300 mg (C13011 Placebo) | Vedolizumab 300 mg (C13011 Vedolizumab) | Vedolizumab 300 mg (C13008 De Novo Participants - UC) | Vedolizumab 300 mg (C13008 De Novo Participants - CD)
Number analyzed (Participants) | 32 | 64 | 69 | 49 | 56 | 63 | 107 | 118 | 133 | 135
score on a scale
  Baseline | 39.33 (11.878) | 41.18 (11.150) | 38.29 (11.062) | 35.43 (11.445) | 39.45 (9.910) | 38.98 (11.963) | 36.80 (11.052) | 38.54 (12.379) | 40.32 (11.333) | 39.16 (11.518)
  Change at Week 52 | 10.27 (12.895) | 10.40 (10.777) | 12.18 (11.506) | 12.68 (11.843) | 10.54 (11.719) | 8.40 (11.598) | 8.27 (11.770) | 7.86 (13.129) | 6.71 (10.363) | 6.23 (12.306)

21. Primary Outcome: Change From Baseline in Short Form-36 (SF-36) Physical Component at Week 76
Description: as for outcome 17
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vedolizumab 300 mg (C13006 Placebo) | Vedolizumab 300 mg (C13006 Vedolizumab Q8W) | Vedolizumab 300 mg (C13006 Vedolizumab Q4W) | Vedolizumab 300 mg (C13007 Placebo) | Vedolizumab 300 mg (C13007 Vedolizumab Q8W) | Vedolizumab 300 mg (C13007 Vedolizumab Q4W) | Vedolizumab 300 mg (C13011 Placebo) | Vedolizumab 300 mg (C13011 Vedolizumab) | Vedolizumab 300 mg (C13008 De Novo Participants - UC) | Vedolizumab 300 mg (C13008 De Novo Participants - CD)
Number analyzed (Participants) | 29 | 63 | 63 | 45 | 55 | 58 | 90 | 106 | 120 | 114
score on a scale
  Baseline | 39.79 (8.801) | 41.33 (8.517) | 40.07 (7.625) | 37.03 (7.675) | 37.92 (8.353) | 39.59 (7.809) | 37.53 (8.286) | 37.47 (8.147) | 40.73 (8.552) | 39.25 (7.667)
  Change at Week 76 | 9.69 (9.714) | 8.97 (8.891) | 10.54 (6.416) | 10.48 (7.797) | 11.98 (9.496) | 10.28 (7.651) | 7.77 (8.397) | 8.82 (8.501) | 9.73 (8.461) | 7.31 (8.436)

22. Primary Outcome: Change From Baseline in Short Form-36 (SF-36) Mental Component Score at Week 76
Description: as for outcome 18
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vedolizumab 300 mg (C13006 Placebo) | Vedolizumab 300 mg (C13006 Vedolizumab Q8W) | Vedolizumab 300 mg (C13006 Vedolizumab Q4W) | Vedolizumab 300 mg (C13007 Placebo) | Vedolizumab 300 mg (C13007 Vedolizumab Q8W) | Vedolizumab 300 mg (C13007 Vedolizumab Q4W) | Vedolizumab 300 mg (C13011 Placebo) | Vedolizumab 300 mg (C13011 Vedolizumab) | Vedolizumab 300 mg (C13008 De Novo Participants - UC) | Vedolizumab 300 mg (C13008 De Novo Participants - CD)
Number analyzed (Participants) | 29 | 63 | 63 | 45 | 55 | 58 | 90 | 106 | 120 | 114
score on a scale
  Baseline | 39.41 (11.201) | 41.30 (10.710) | 38.26 (10.974) | 35.50 (11.582) | 38.86 (10.046) | 38.52 (12.244) | 36.68 (11.947) | 39.03 (12.679) | 40.32 (11.673) | 39.16 (11.712)
  Change at Week 76 | 9.64 (14.272) | 8.52 (11.462) | 10.51 (12.334) | 12.92 (13.174) | 8.02 (14.020) | 9.13 (13.719) | 8.27 (12.720) | 8.26 (12.809) | 7.77 (10.989) | 7.16 (13.144)

23. Primary Outcome: Change From Baseline in Short Form-36 (SF-36) Physical Component Score at Week 100
Description: as for outcome 17
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vedolizumab 300 mg (C13006 Placebo) | Vedolizumab 300 mg (C13006 Vedolizumab Q8W) | Vedolizumab 300 mg (C13006 Vedolizumab Q4W) | Vedolizumab 300 mg (C13007 Placebo) | Vedolizumab 300 mg (C13007 Vedolizumab Q8W) | Vedolizumab 300 mg (C13007 Vedolizumab Q4W) | Vedolizumab 300 mg (C13011 Placebo) | Vedolizumab 300 mg (C13011 Vedolizumab) | Vedolizumab 300 mg (C13008 De Novo Participants - UC) | Vedolizumab 300 mg (C13008 De Novo Participants - CD)
Number analyzed (Participants) | 27 | 58 | 58 | 45 | 49 | 54 | 84 | 96 | 114 | 105
score on a scale
  Baseline | 41.26 (8.825) | 41.03 (8.260) | 40.29 (7.480) | 36.97 (7.677) | 38.11 (8.169) | 39.59 (7.989) | 37.26 (7.974) | 37.90 (8.297) | 41.13 (8.579) | 39.28 (7.458)
  Change at Week 100 | 10.28 (8.418) | 9.41 (7.934) | 9.42 (7.556) | 11.18 (8.322) | 12.97 (9.396) | 10.78 (8.926) | 8.47 (8.096) | 9.45 (8.747) | 9.70 (8.869) | 7.40 (8.473)

24. Primary Outcome: Change From Baseline in Short Form-36 (SF-36) Mental Component Score at Week 100
Description: as for outcome 18
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vedolizumab 300 mg (C13006 Placebo) | Vedolizumab 300 mg (C13006 Vedolizumab Q8W) | Vedolizumab 300 mg (C13006 Vedolizumab Q4W) | Vedolizumab 300 mg (C13007 Placebo) | Vedolizumab 300 mg (C13007 Vedolizumab Q8W) | Vedolizumab 300 mg (C13007 Vedolizumab Q4W) | Vedolizumab 300 mg (C13011 Placebo) | Vedolizumab 300 mg (C13011 Vedolizumab) | Vedolizumab 300 mg (C13008 De Novo Participants - UC) | Vedolizumab 300 mg (C13008 De Novo Participants - CD)
Number analyzed (Participants) | 27 | 58 | 58 | 45 | 49 | 54 | 84 | 96 | 114 | 105
score on a scale
  Baseline | 39.56 (11.833) | 41.10 (11.140) | 38.21 (10.885) | 35.61 (11.568) | 38.76 (10.215) | 37.41 (11.857) | 36.61 (11.894) | 39.43 (12.474) | 40.39 (11.559) | 39.04 (11.604)
  Change at Week 100 | 8.80 (14.395) | 9.87 (10.552) | 10.82 (12.303) | 10.64 (13.629) | 8.94 (13.798) | 9.98 (11.450) | 8.25 (12.562) | 7.93 (11.053) | 7.66 (10.685) | 6.94 (13.189)

25. Primary Outcome: Change From Baseline in Short Form-36 (SF-36) Physical Component Scores at Week 124
Description: as for outcome 17
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vedolizumab 300 mg (C13006 Placebo) | Vedolizumab 300 mg (C13006 Vedolizumab Q8W) | Vedolizumab 300 mg (C13006 Vedolizumab Q4W) | Vedolizumab 300 mg (C13007 Placebo) | Vedolizumab 300 mg (C13007 Vedolizumab Q8W) | Vedolizumab 300 mg (C13007 Vedolizumab Q4W) | Vedolizumab 300 mg (C13011 Placebo) | Vedolizumab 300 mg (C13011 Vedolizumab) | Vedolizumab 300 mg (C13008 De Novo Participants - UC) | Vedolizumab 300 mg (C13008 De Novo Participants - CD)
Number analyzed (Participants) | 27 | 58 | 54 | 43 | 47 | 48 | 80 | 83 | 97 | 98
score on a scale
  Baseline | 41.75 (7.947) | 41.08 (8.219) | 39.88 (7.332) | 37.00 (7.854) | 38.58 (8.078) | 39.31 (8.279) | 37.09 (8.044) | 38.36 (8.240) | 41.10 (8.747) | 39.01 (7.363)
  Change at Week 124 | 10.12 (9.685) | 7.91 (9.483) | 10.15 (8.551) | 11.79 (8.053) | 12.87 (8.803) | 11.01 (8.319) | 8.36 (7.495) | 7.77 (9.228) | 10.56 (8.804) | 9.27 (8.274)

26. Primary Outcome: Change From Baseline in Short Form-36 (SF-36) Mental Component Scores at Week 124
Description: as for outcome 18
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vedolizumab 300 mg (C13006 Placebo) | Vedolizumab 300 mg (C13006 Vedolizumab Q8W) | Vedolizumab 300 mg (C13006 Vedolizumab Q4W) | Vedolizumab 300 mg (C13007 Placebo) | Vedolizumab 300 mg (C13007 Vedolizumab Q8W) | Vedolizumab 300 mg (C13007 Vedolizumab Q4W) | Vedolizumab 300 mg (C13011 Placebo) | Vedolizumab 300 mg (C13011 Vedolizumab) | Vedolizumab 300 mg (C13008 De Novo Participants - UC) | Vedolizumab 300 mg (C13008 De Novo Participants - CD)
Number analyzed (Participants) | 27 | 58 | 54 | 43 | 47 | 48 | 80 | 83 | 97 | 98
score on a scale
  Baseline | 40.34 (12.065) | 40.81 (11.132) | 37.85 (11.106) | 35.29 (11.668) | 38.59 (9.956) | 38.33 (12.409) | 39.04 (12.421) | 36.64 (11.938) | 40.87 (11.156) | 38.90 (11.427)
  Change at Week 124 | 9.53 (16.289) | 10.02 (10.734) | 9.70 (12.781) | 11.35 (12.681) | 9.20 (12.521) | 10.38 (13.230) | 8.50 (12.808) | 8.78 (13.283) | 7.73 (11.048) | 6.26 (13.274)

27. Primary Outcome: Change From Baseline in Short Form-36 (SF-36) Physical Component Score at Week 148
Description: The Short Form-36 (SF-36) is a questionnaire that evaluates a person's HRQOL. SF-36 includes 36 questions related to 8 health dimensions: physical functioning, role-physical (role limitations due to physical health problems), bodily pain, general health, vitality (energy/fatigue), social functioning, role-emotional (role limitations due to emotional problems), and mental health. Based on these 8 scales, the physical component summary (PCS) score is generated which ranges between 0 and 100, with higher scores indicating a better quality of life. A positive change from Baseline indicates improvement.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vedolizumab 300 mg (C13006 Placebo) | Vedolizumab 300 mg (C13006 Vedolizumab Q8W) | Vedolizumab 300 mg (C13006 Vedolizumab Q4W) | Vedolizumab 300 mg (C13007 Placebo) | Vedolizumab 300 mg (C13007 Vedolizumab Q8W) | Vedolizumab 300 mg (C13007 Vedolizumab Q4W) | Vedolizumab 300 mg (C13011 Placebo) | Vedolizumab 300 mg (C13011 Vedolizumab) | Vedolizumab 300 mg (C13008 De Novo Participants - UC) | Vedolizumab 300 mg (C13008 De Novo Participants - CD)
Number analyzed (Participants) | 27 | 58 | 53 | 40 | 43 | 46 | 76 | 82 | 20 | 24
score on a scale
  Baseline | 41.75 (7.947) | 41.33 (8.438) | 39.86 (7.312) | 36.68 (8.055) | 39.22 (7.511) | 39.21 (8.303) | 36.94 (8.087) | 37.99 (8.430) | 43.32 (10.405) | 38.77 (7.024)
  Change at Week 148 | 9.08 (9.090) | 9.35 (8.228) | 10.34 (6.524) | 12.15 (9.941) | 12.54 (9.695) | 11.26 (7.231) | 9.37 (8.223) | 8.94 (8.442) | 9.81 (8.727) | 10.39 (6.824)

28. Primary Outcome: Change From Baseline in Short Form-36 (SF-36) Mental Component Score at Week 148
Description: as for outcome 18
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vedolizumab 300 mg (C13006 Placebo) | Vedolizumab 300 mg (C13006 Vedolizumab Q8W) | Vedolizumab 300 mg (C13006 Vedolizumab Q4W) | Vedolizumab 300 mg (C13007 Placebo) | Vedolizumab 300 mg (C13007 Vedolizumab Q8W) | Vedolizumab 300 mg (C13007 Vedolizumab Q4W) | Vedolizumab 300 mg (C13011 Placebo) | Vedolizumab 300 mg (C13011 Vedolizumab) | Vedolizumab 300 mg (C13008 De Novo Participants - UC) | Vedolizumab 300 mg (C13008 De Novo Participants - CD)
Number analyzed (Participants) | 27 | 54 | 53 | 40 | 43 | 46 | 76 | 82 | 20 | 24
score on a scale
  Baseline | 40.34 (12.065) | 41.20 (11.115) | 37.48 (11.101) | 35.05 (11.782) | 38.56 (10.221) | 39.21 (12.368) | 36.71 (12.021) | 39.36 (12.612) | 42.40 (8.427) | 41.67 (10.953)
  Change at Week 148 | 6.89 (14.522) | 9.79 (11.176) | 11.09 (12.299) | 10.47 (12.517) | 9.27 (11.720) | 9.81 (12.524) | 8.91 (12.680) | 8.26 (12.835) | 6.44 (12.279) | 6.85 (12.118)

29. Primary Outcome: Change From Baseline in Short Form-36 (SF-36) Physical Component Scores at Week 172
Description: as for outcome 17
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vedolizumab 300 mg (C13006 Placebo) | Vedolizumab 300 mg (C13006 Vedolizumab Q8W) | Vedolizumab 300 mg (C13006 Vedolizumab Q4W) | Vedolizumab 300 mg (C13007 Placebo) | Vedolizumab 300 mg (C13007 Vedolizumab Q8W) | Vedolizumab 300 mg (C13007 Vedolizumab Q4W) | Vedolizumab 300 mg (C13011 Placebo) | Vedolizumab 300 mg (C13011 Vedolizumab) | Vedolizumab 300 mg (C13008 De Novo Participants - UC) | Vedolizumab 300 mg (C13008 De Novo Participants - CD)
Number analyzed (Participants) | 25 | 53 | 49 | 37 | 43 | 43 | 71 | 75 | 91 | 81
score on a scale
  Baseline | 42.23 (8.073) | 41.52 (8.401) | 40.23 (6.713) | 37.29 (8.057) | 38.82 (8.231) | 39.16 (8.177) | 36.92 (8.023) | 37.85 (8.538) | 41.12 (9.029) | 39.30 (7.264)
  Change at Week 172 | 10.08 (8.996) | 9.20 (8.324) | 9.68 (6.804) | 11.83 (8.042) | 13.21 (9.194) | 10.88 (7.837) | 9.61 (8.461) | 9.07 (7.519) | 10.47 (8.921) | 8.55 (8.546)

30. Primary Outcome: Change From Baseline in Short Form-36 (SF-36) Mental Component Scores at Week 172
Description: as for outcome 18
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vedolizumab 300 mg (C13006 Placebo) | Vedolizumab 300 mg (C13006 Vedolizumab Q8W) | Vedolizumab 300 mg (C13006 Vedolizumab Q4W) | Vedolizumab 300 mg (C13007 Placebo) | Vedolizumab 300 mg (C13007 Vedolizumab Q8W) | Vedolizumab 300 mg (C13007 Vedolizumab Q4W) | Vedolizumab 300 mg (C13011 Placebo) | Vedolizumab 300 mg (C13011 Vedolizumab) | Vedolizumab 300 mg (C13008 De Novo Participants - UC) | Vedolizumab 300 mg (C13008 De Novo Participants - CD)
Number analyzed (Participants) | 25 | 53 | 49 | 37 | 43 | 43 | 71 | 75 | 91 | 81
score on a scale
  Baseline | 40.79 (12.254) | 41.49 (11.015) | 37.00 (10.963) | 35.47 (11.757) | 38.77 (10.268) | 39.83 (12.249) | 36.64 (11.938) | 39.01 (12.258) | 40.98 (11.479) | 38.85 (11.972)
  Change at Week 172 | 7.43 (12.227) | 10.37 (10.420) | 9.57 (12.850) | 12.84 (12.281) | 9.12 (14.244) | 8.45 (13.317) | 8.78 (13.283) | 7.52 (12.609) | 8.66 (10.767) | 7.48 (12.329)

31. Primary Outcome: Change From Baseline in Short Form-36 (SF-36) Physical Component Score at Week 196
Description: as for outcome 17
Time Frame: as for outcome 13
Population: ITT population from studies C13006, C13007 and C13011 who received vedolizumab in study C13008. Data is provided for participants who were completers in previous studies with data available at both Baseline and Week 196. Not applicable for Vedolizumab 300 mg (C13004) arm group. Data is not available for de novo participants at this time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vedolizumab 300 mg (C13006 Placebo) | Vedolizumab 300 mg (C13006 Vedolizumab Q8W) | Vedolizumab 300 mg (C13006 Vedolizumab Q4W) | Vedolizumab 300 mg (C13007 Placebo) | Vedolizumab 300 mg (C13007 Vedolizumab Q8W) | Vedolizumab 300 mg (C13007 Vedolizumab Q4W) | Vedolizumab 300 mg (C13011 Placebo) | Vedolizumab 300 mg (C13011 Vedolizumab)
Number analyzed (Participants) | 16 | 33 | 29 | 31 | 27 | 33 | 19 | 21
score on a scale
  Baseline | 40.72 (7.823) | 40.83 (8.135) | 40.52 (7.242) | 35.64 (7.862) | 36.65 (9.250) | 39.33 (8.136) | 39.53 (7.830) | 38.40 (9.680)
  Change at Week 196 | 11.82 (9.370) | 9.98 (7.569) | 9.31 (5.771) | 12.35 (8.867) | 14.10 (10.616) | 11.75 (8.261) | 6.94 (8.667) | 9.83 (8.111)

32. Primary Outcome: Change From Baseline in Short Form-36 (SF-36) Mental Component Score at Week 196
Description: as for outcome 18
Time Frame: as for outcome 13
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vedolizumab 300 mg (C13006 Placebo) | Vedolizumab 300 mg (C13006 Vedolizumab Q8W) | Vedolizumab 300 mg (C13006 Vedolizumab Q4W) | Vedolizumab 300 mg (C13007 Placebo) | Vedolizumab 300 mg (C13007 Vedolizumab Q8W) | Vedolizumab 300 mg (C13007 Vedolizumab Q4W) | Vedolizumab 300 mg (C13011 Placebo) | Vedolizumab 300 mg (C13011 Vedolizumab)
Number analyzed (Participants) | 16 | 33 | 29 | 31 | 27 | 33 | 19 | 21
score on a scale
  Baseline | 39.46 (13.424) | 42.74 (10.517) | 40.40 (9.771) | 36.17 (12.536) | 39.07 (10.804) | 37.63 (12.199) | 40.11 (10.932) | 40.05 (13.807)
  Change at Week 196 | 9.37 (12.087) | 9.43 (9.349) | 9.79 (11.516) | 12.62 (14.386) | 10.05 (15.471) | 9.26 (12.732) | 8.59 (14.645) | 9.75 (14.824)

33. Primary Outcome: Change From Baseline in Short Form-36 (SF-36) Physical Component Score at Week 248
Description: as for outcome 17
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vedolizumab 300 mg (C13006 Placebo) | Vedolizumab 300 mg (C13006 Vedolizumab Q8W) | Vedolizumab 300 mg (C13006 Vedolizumab Q4W) | Vedolizumab 300 mg (C13007 Placebo) | Vedolizumab 300 mg (C13007 Vedolizumab Q8W) | Vedolizumab 300 mg (C13007 Vedolizumab Q4W) | Vedolizumab 300 mg (C13011 Placebo) | Vedolizumab 300 mg (C13011 Vedolizumab) | Vedolizumab 300 mg (C13008 De Novo Participants - UC) | Vedolizumab 300 mg (C13008 De Novo Participants - CD)
Number analyzed (Participants) | 21 | 38 | 36 | 32 | 32 | 31 | 38 | 45 | 3 | 4
score on a scale
  Baseline | 39.99 (7.219) | 40.71 (7.605) | 39.33 (6.820) | 37.54 (8.054) | 38.32 (8.047) | 40.28 (8.878) | 37.95 (8.232) | 37.77 (8.654) | 39.17 (13.987) | 38.79 (7.735)
  Change at Week 248 | 11.22 (10.562) | 9.95 (8.355) | 11.43 (8.047) | 11.70 (6.541) | 13.88 (8.511) | 9.98 (9.027) | 9.32 (9.261) | 10.50 (8.803) | 15.98 (7.868) | 9.88 (6.977)

34. Primary Outcome: Change From Baseline in Short Form-36 (SF-36) Mental Component Score at Week 248
Description: as for outcome 18
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vedolizumab 300 mg (C13006 Placebo) | Vedolizumab 300 mg (C13006 Vedolizumab Q8W) | Vedolizumab 300 mg (C13006 Vedolizumab Q4W) | Vedolizumab 300 mg (C13007 Placebo) | Vedolizumab 300 mg (C13007 Vedolizumab Q8W) | Vedolizumab 300 mg (C13007 Vedolizumab Q4W) | Vedolizumab 300 mg (C13011 Placebo) | Vedolizumab 300 mg (C13011 Vedolizumab) | Vedolizumab 300 mg (C13008 De Novo Participants - UC) | Vedolizumab 300 mg (C13008 De Novo Participants - CD)
Number analyzed (Participants) | 21 | 38 | 36 | 32 | 32 | 31 | 38 | 45 | 3 | 4
score on a scale
  Baseline | 38.00 (12.537) | 41.76 (10.579) | 38.01 (10.876) | 34.26 (12.252) | 38.06 (10.300) | 38.04 (11.320) | 36.41 (13.568) | 36.77 (12.333) | 38.65 (18.372) | 31.20 (4.603)
  Change at Week 248 | 11.99 (13.421) | 6.13 (9.986) | 10.41 (13.081) | 12.70 (12.140) | 9.84 (11.433) | 10.61 (11.204) | 7.37 (16.473) | 10.61 (12.188) | 7.64 (18.599) | 15.98 (13.355)

35. Primary Outcome: Change From Baseline in Short Form-36 (SF-36) Physical Component Score at Week 300
Description: as for outcome 17
Time Frame: as for outcome 15
Population: ITT population from studies C13006, C13007 and C13011 who received vedolizumab in study C13008. Data is provided for participants who were completers in previous studies with data available at both Baseline and Week 300. Not applicable for Vedolizumab 300 mg (C13004) arm group. Data is not available for de novo participants at this time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vedolizumab 300 mg (C13006 Placebo) | Vedolizumab 300 mg (C13006 Vedolizumab Q8W) | Vedolizumab 300 mg (C13006 Vedolizumab Q4W) | Vedolizumab 300 mg (C13007 Placebo) | Vedolizumab 300 mg (C13007 Vedolizumab Q8W) | Vedolizumab 300 mg (C13007 Vedolizumab Q4W) | Vedolizumab 300 mg (C13011 Placebo) | Vedolizumab 300 mg (C13011 Vedolizumab)
Number analyzed (Participants) | 7 | 14 | 13 | 9 | 8 | 16 | 4 | 2
score on a scale
  Baseline | 36.89 (5.913) | 38.84 (7.720) | 39.22 (5.469) | 36.56 (8.514) | 34.80 (8.431) | 39.97 (6.626) | 41.04 (12.016) | 34.80 (10.515)
  Change at Week 300 | 12.03 (10.338) | 10.58 (8.335) | 11.15 (6.497) | 15.47 (9.920) | 14.42 (6.749) | 10.69 (6.448) | 9.10 (9.330) | 6.41 (9.023)

36. Primary Outcome: Change From Baseline in Short Form-36 (SF-36) Mental Component Score at Week 300
Description: as for outcome 18
Time Frame: as for outcome 15
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vedolizumab 300 mg (C13006 Placebo) | Vedolizumab 300 mg (C13006 Vedolizumab Q8W) | Vedolizumab 300 mg (C13006 Vedolizumab Q4W) | Vedolizumab 300 mg (C13007 Placebo) | Vedolizumab 300 mg (C13007 Vedolizumab Q8W) | Vedolizumab 300 mg (C13007 Vedolizumab Q4W) | Vedolizumab 300 mg (C13011 Placebo) | Vedolizumab 300 mg (C13011 Vedolizumab)
Number analyzed (Participants) | 7 | 14 | 13 | 9 | 8 | 16 | 4 | 2
score on a scale
  Baseline | 34.53 (12.530) | 43.55 (9.074) | 35.77 (8.585) | 33.38 (11.168) | 39.40 (11.144) | 35.79 (12.157) | 31.35 (13.760) | 46.99 (7.729)
  Change at Week 300 | 21.86 (13.935) | 4.82 (10.738) | 9.82 (11.463) | 13.46 (15.324) | 6.31 (11.916) | 14.79 (15.281) | 19.87 (6.588) | -3.67 (20.577)

37. Primary Outcome: Change From Baseline in Short Form-36 (SF-36) Physical Component Score at Week 352
Description: as for outcome 27
Time Frame: as for outcome 16
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vedolizumab 300 mg (C13006 Placebo) | Vedolizumab 300 mg (C13006 Vedolizumab Q8W) | Vedolizumab 300 mg (C13006 Vedolizumab Q4W) | Vedolizumab 300 mg (C13007 Placebo) | Vedolizumab 300 mg (C13007 Vedolizumab Q8W) | Vedolizumab 300 mg (C13007 Vedolizumab Q4W)
Number analyzed (Participants) | 1 | 1 | 3 | 1 | 2 | 1
score on a scale
  Baseline | 35.68 (NA) — SD was not calculated for 1 participant. | 38.32 (NA) — SD was not calculated for 1 participant. | 44.36 (0.920) | 31.07 (NA) — SD was not calculated for 1 participant. | 37.14 (3.711) | 33.67 (NA) — SD was not calculated for 1 participant.
  Change at Week 352 | 17.97 (NA) — SD was not calculated for 1 participant. | 17.87 (NA) — SD was not calculated for 1 participant. | 5.06 (5.188) | 24.06 (NA) — SD was not calculated for 1 participant. | 11.18 (2.116) | 18.02 (NA) — SD was not calculated for 1 participant.

38. Primary Outcome: Change From Baseline in Short Form-36 (SF-36) Mental Component Score at Week 352
Description: as for outcome 18
Time Frame: as for outcome 16
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vedolizumab 300 mg (C13006 Placebo) | Vedolizumab 300 mg (C13006 Vedolizumab Q8W) | Vedolizumab 300 mg (C13006 Vedolizumab Q4W) | Vedolizumab 300 mg (C13007 Placebo) | Vedolizumab 300 mg (C13007 Vedolizumab Q8W) | Vedolizumab 300 mg (C13007 Vedolizumab Q4W)
Number analyzed (Participants) | 1 | 1 | 3 | 1 | 2 | 1
score on a scale
  Baseline | 42.19 (NA) — SD was not calculated for 1 participant. | 35.34 (NA) — SD was not calculated for 1 participant. | 32.72 (7.252) | 22.18 (NA) — SD was not calculated for 1 participant. | 39.80 (14.563) | 42.98 (NA) — SD was not calculated for 1 participant.
  Change at Week 352 | 17.40 (NA) — SD was not calculated for 1 participant. | 19.87 (NA) — SD was not calculated for 1 participant. | 14.14 (10.114) | 25.04 (NA) — SD was not calculated for 1 participant. | 8.65 (7.463) | 13.08 (NA) — SD was not calculated for 1 participant.

39. Primary Outcome: Change From Baseline in European Quality of Life 5-Dimension (EQ-5D) Health States Composite Score at Week 28
Description: EQ-5D health states questionnaire is an instrument used to measure general health related quality of life (HRQOL) in participants with infectious bowel disease (IBD). It considers five attributes of quality of life evaluation: mobility, self-care, usual activity, pain/discomfort, and anxiety/depression. Each dimension has three possible levels: 1=none, 2=moderate or 3=extreme. A composite EQ-5D score can be calculated from the individual scores to assess overall HRQOL. A composite EQ-5D score is calculated as a sum of all 5 sub-scores. The total sub-score ranges from 5 to 15. A decrease of ≥0.3 points in the composite EQ-5D score represents improvement in quality of life of participants. A negative change from Baseline indicates improvement.
Time Frame: as for outcome 6
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vedolizumab 300 mg (C13006 Placebo) | Vedolizumab 300 mg (C13006 Vedolizumab Q8W) | Vedolizumab 300 mg (C13006 Vedolizumab Q4W) | Vedolizumab 300 mg (C13007 Placebo) | Vedolizumab 300 mg (C13007 Vedolizumab Q8W) | Vedolizumab 300 mg (C13007 Vedolizumab Q4W) | Vedolizumab 300 mg (C13011 Placebo) | Vedolizumab 300 mg (C13011 Vedolizumab) | Vedolizumab 300 mg (C13008 De Novo Participants - UC) | Vedolizumab 300 mg (C13008 De Novo Participants - CD)
Number analyzed (Participants) | 38 | 67 | 76 | 52 | 62 | 71 | 126 | 136 | 151 | 162
score on a scale
  Baseline | 7.42 (1.328) | 7.21 (1.354) | 7.54 (1.399) | 8.00 (1.559) | 7.77 (1.442) | 7.73 (1.434) | 7.67 (1.475) | 7.85 (1.525) | 7.30 (1.360) | 7.48 (1.420)
  Change at Week 28 | -1.29 (1.873) | -1.03 (1.705) | -1.44 (1.568) | -1.65 (1.867) | -1.82 (1.675) | -1.46 (1.510) | -0.75 (1.648) | -0.90 (1.634) | -0.96 (1.380) | -0.69 (1.493)

40. Primary Outcome: Change From Baseline in European Quality of Life 5-Dimension (EQ-5D) Health States Visual Analog Scale (VAS) Score at Week 28
Description: EQ-5D questionnaire is an instrument used to measure general HRQOL in participants with IBD. Each dimension has three possible levels: 1 = none, 2 = moderate or 3 = extreme. The EQ-5D VAS score is a self-assigned rating of overall health using a 20-cm visual, vertical scale, with a score of 0 as the worst and 100 as the best possible health. An increase of ≥7 points in the EQ-5D VAS score represents a clinically meaningful improvement in quality of life for participants. A positive change from Baseline indicates improvement.
Time Frame: as for outcome 6
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vedolizumab 300 mg (C13006 Placebo) | Vedolizumab 300 mg (C13006 Vedolizumab Q8W) | Vedolizumab 300 mg (C13006 Vedolizumab Q4W) | Vedolizumab 300 mg (C13007 Placebo) | Vedolizumab 300 mg (C13007 Vedolizumab Q8W) | Vedolizumab 300 mg (C13007 Vedolizumab Q4W) | Vedolizumab 300 mg (C13011 Placebo) | Vedolizumab 300 mg (C13011 Vedolizumab) | Vedolizumab 300 mg (C13008 De Novo Participants - UC) | Vedolizumab 300 mg (C13008 De Novo Participants - CD)
Number analyzed (Participants) | 38 | 67 | 75 | 52 | 62 | 70 | 125 | 135 | 149 | 157
score on a scale
  Baseline | 58.4 (20.96) | 62.1 (16.54) | 53.5 (17.30) | 51.5 (17.57) | 52.2 (18.72) | 52.3 (18.39) | 53.2 (18.02) | 51.3 (19.09) | 56.4 (19.64) | 55.6 (16.72)
  Change at Week 28 | 22.7 (24.11) | 20.0 (18.75) | 25.1 (22.09) | 23.8 (23.79) | 27.6 (22.58) | 23.7 (22.51) | 16.8 (22.55) | 19.9 (22.44) | 17.1 (21.75) | 13.4 (19.48)

41. Primary Outcome: Change From Baseline in European Quality of Life 5-Dimension (EQ-5D) Health States Composite Score at Week 52
Description: as for outcome 39
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vedolizumab 300 mg (C13006 Placebo) | Vedolizumab 300 mg (C13006 Vedolizumab Q8W) | Vedolizumab 300 mg (C13006 Vedolizumab Q4W) | Vedolizumab 300 mg (C13007 Placebo) | Vedolizumab 300 mg (C13007 Vedolizumab Q8W) | Vedolizumab 300 mg (C13007 Vedolizumab Q4W) | Vedolizumab 300 mg (C13011 Placebo) | Vedolizumab 300 mg (C13011 Vedolizumab) | Vedolizumab 300 mg (C13008 De Novo Participants - UC) | Vedolizumab 300 mg (C13008 De Novo Participants - CD)
Number analyzed (Participants) | 32 | 65 | 70 | 48 | 56 | 63 | 107 | 118 | 133 | 135
score on a scale
  Baseline | 7.50 (1.368) | 7.17 (1.318) | 7.54 (1.390) | 8.08 (1.499) | 7.75 (1.468) | 7.65 (1.358) | 7.62 (1.398) | 7.74 (1.538) | 7.33 (1.386) | 7.49 (1.429)
  Change at Week 52 | -1.59 (1.775) | -1.00 (1.571) | -1.43 (1.556) | -1.60 (1.673) | -1.77 (1.640) | -1.46 (1.457) | -0.87 (1.666) | -1.15 (1.703) | -0.95 (1.551) | -0.85 (1.637)

42. Primary Outcome: Change From Baseline in European Quality of Life 5-Dimension (EQ-5D) Health States Visual Analog Scale (VAS) Score at Week 52
Description: as for outcome 40
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vedolizumab 300 mg (C13006 Placebo) | Vedolizumab 300 mg (C13006 Vedolizumab Q8W) | Vedolizumab 300 mg (C13006 Vedolizumab Q4W) | Vedolizumab 300 mg (C13007 Placebo) | Vedolizumab 300 mg (C13007 Vedolizumab Q8W) | Vedolizumab 300 mg (C13007 Vedolizumab Q4W) | Vedolizumab 300 mg (C13011 Placebo) | Vedolizumab 300 mg (C13011 Vedolizumab) | Vedolizumab 300 mg (C13008 De Novo Participants - UC) | Vedolizumab 300 mg (C13008 De Novo Participants - CD)
Number analyzed (Participants) | 31 | 65 | 70 | 49 | 56 | 62 | 105 | 118 | 129 | 133
score on a scale
  Baseline | 57.5 (21.39) | 61.9 (16.18) | 52.3 (18.09) | 50.8 (17.82) | 52.6 (19.43) | 52.7 (18.38) | 53.3 (17.21) | 52.2 (18.94) | 55.9 (20.51) | 56.3 (16.21)
  Change at Week 52 | 22.9 (27.46) | 18.5 (20.31) | 27.0 (21.87) | 27.9 (20.70) | 30.8 (21.59) | 25.0 (18.85) | 19.9 (22.83) | 23.5 (23.03) | 20.8 (21.93) | 17.6 (22.69)

43. Primary Outcome: Change From Baseline in European Quality of Life 5-Dimension (EQ-5D) Health States Composite Score at Week 76
Description: as for outcome 39
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vedolizumab 300 mg (C13006 Placebo) | Vedolizumab 300 mg (C13006 Vedolizumab Q8W) | Vedolizumab 300 mg (C13006 Vedolizumab Q4W) | Vedolizumab 300 mg (C13007 Placebo) | Vedolizumab 300 mg (C13007 Vedolizumab Q8W) | Vedolizumab 300 mg (C13007 Vedolizumab Q4W) | Vedolizumab 300 mg (C13011 Placebo) | Vedolizumab 300 mg (C13011 Vedolizumab) | Vedolizumab 300 mg (C13008 De Novo Participants - UC) | Vedolizumab 300 mg (C13008 De Novo Participants - CD)
Number analyzed (Participants) | 29 | 62 | 63 | 45 | 54 | 58 | 89 | 106 | 120 | 113
score on a scale
  Baseline | 7.48 (1.379) | 7.18 (1.337) | 7.56 (1.267) | 8.11 (1.434) | 7.72 (1.420) | 7.64 (1.385) | 7.69 (1.489) | 7.74 (1.545) | 7.28 (1.348) | 7.52 (1.464)
  Change at Week 76 | -1.38 (1.498) | -1.05 (1.583) | -1.33 (1.513) | -1.67 (1.430) | -1.50 (1.724) | -1.52 (1.466) | -1.11 (1.518) | -1.14 (1.496) | -1.26 (1.481) | -1.05 (1.546)

44. Primary Outcome: Change From Baseline in European Quality of Life 5-Dimension (EQ-5D) Health States Visual Analog Scale (VAS) Score at Week 76
Description: as for outcome 40
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vedolizumab 300 mg (C13006 Placebo) | Vedolizumab 300 mg (C13006 Vedolizumab Q8W) | Vedolizumab 300 mg (C13006 Vedolizumab Q4W) | Vedolizumab 300 mg (C13007 Placebo) | Vedolizumab 300 mg (C13007 Vedolizumab Q8W) | Vedolizumab 300 mg (C13007 Vedolizumab Q4W) | Vedolizumab 300 mg (C13011 Placebo) | Vedolizumab 300 mg (C13011 Vedolizumab) | Vedolizumab 300 mg (C13008 De Novo Participants - UC) | Vedolizumab 300 mg (C13008 De Novo Participants - CD)
Number analyzed (Participants) | 29 | 62 | 63 | 44 | 54 | 57 | 88 | 106 | 119 | 113
score on a scale
  Baseline | 58.8 (21.93) | 62.3 (17.01) | 52.0 (18.47) | 50.7 (16.81) | 52.0 (19.38) | 52.4 (18.88) | 52.5 (17.18) | 51.4 (18.99) | 56.1 (20.36) | 55.8 (16.19)
  Change at Week 76 | 20.9 (25.66) | 18.7 (20.65) | 25.1 (19.62) | 27.3 (18.87) | 30.3 (23.68) | 27.0 (21.49) | 22.2 (20.82) | 23.3 (21.40) | 19.2 (25.10) | 17.8 (22.04)

45. Primary Outcome: Change From Baseline in European Quality of Life 5-Dimension (EQ-5D) Health States Composite Score at Week 100
Description: as for outcome 39
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vedolizumab 300 mg (C13006 Placebo) | Vedolizumab 300 mg (C13006 Vedolizumab Q8W) | Vedolizumab 300 mg (C13006 Vedolizumab Q4W) | Vedolizumab 300 mg (C13007 Placebo) | Vedolizumab 300 mg (C13007 Vedolizumab Q8W) | Vedolizumab 300 mg (C13007 Vedolizumab Q4W) | Vedolizumab 300 mg (C13011 Placebo) | Vedolizumab 300 mg (C13011 Vedolizumab) | Vedolizumab 300 mg (C13008 De Novo Participants - UC) | Vedolizumab 300 mg (C13008 De Novo Participants - CD)
Number analyzed (Participants) | 27 | 58 | 58 | 45 | 49 | 55 | 84 | 96 | 114 | 105
score on a scale
  Baseline | 7.48 (1.451) | 7.22 (1.325) | 7.55 (1.391) | 8.04 (1.507) | 7.69 (1.446) | 7.67 (1.375) | 7.71 (1.428) | 7.71 (1.507) | 7.28 (1.360) | 7.53 (1.401)
  Change at Week 100 | -1.48 (1.602) | -1.26 (1.528) | -1.43 (1.452) | -1.64 (1.773) | -1.73 (1.741) | -1.62 (1.394) | -1.04 (1.609) | -1.16 (1.538) | -1.37 (1.477) | -0.98 (1.473)

46. Primary Outcome: Change From Baseline in European Quality of Life 5-Dimension (EQ-5D) Health States Visual Analog Scale (VAS) Score at Week 100
Description: as for outcome 40
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vedolizumab 300 mg (C13006 Placebo) | Vedolizumab 300 mg (C13006 Vedolizumab Q8W) | Vedolizumab 300 mg (C13006 Vedolizumab Q4W) | Vedolizumab 300 mg (C13007 Placebo) | Vedolizumab 300 mg (C13007 Vedolizumab Q8W) | Vedolizumab 300 mg (C13007 Vedolizumab Q4W) | Vedolizumab 300 mg (C13011 Placebo) | Vedolizumab 300 mg (C13011 Vedolizumab) | Vedolizumab 300 mg (C13008 De Novo Participants - UC) | Vedolizumab 300 mg (C13008 De Novo Participants - CD)
Number analyzed (Participants) | 27 | 58 | 58 | 44 | 49 | 54 | 82 | 95 | 112 | 103
score on a scale
  Baseline | 59.2 (22.81) | 61.3 (16.80) | 52.9 (16.94) | 50.7 (16.81) | 53.8 (18.76) | 51.9 (19.02) | 51.9 (16.53) | 52.2 (19.18) | 56.5 (20.68) | 55.3 (16.49)
  Change at Week 100 | 20.4 (27.47) | 20.7 (17.45) | 26.4 (21.82) | 26.9 (22.39) | 29.4 (23.09) | 26.9 (21.76) | 22.3 (20.11) | 23.1 (21.82) | 19.4 (26.78) | 16.6 (21.92)

47. Primary Outcome: Change From Baseline in European Quality of Life 5-Dimension (EQ-5D) Health States Composite Score at Week 124
Description: as for outcome 39
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vedolizumab 300 mg (C13006 Placebo) | Vedolizumab 300 mg (C13006 Vedolizumab Q8W) | Vedolizumab 300 mg (C13006 Vedolizumab Q4W) | Vedolizumab 300 mg (C13007 Placebo) | Vedolizumab 300 mg (C13007 Vedolizumab Q8W) | Vedolizumab 300 mg (C13007 Vedolizumab Q4W) | Vedolizumab 300 mg (C13011 Placebo) | Vedolizumab 300 mg (C13011 Vedolizumab) | Vedolizumab 300 mg (C13008 De Novo Participants - UC) | Vedolizumab 300 mg (C13008 De Novo Participants - CD)
Number analyzed (Participants) | 27 | 58 | 54 | 43 | 47 | 48 | 80 | 83 | 97 | 98
score on a scale
  Baseline | 7.33 (1.271) | 7.24 (1.329) | 7.61 (1.406) | 8.14 (1.457) | 7.62 (1.423) | 7.69 (1.446) | 7.73 (1.441) | 7.65 (1.510) | 7.28 (1.223) | 7.54 (1.401)
  Change at Week 124 | -1.52 (1.805) | -1.07 (1.566) | -1.52 (1.539) | -1.70 (1.655) | -1.60 (1.690) | -1.69 (1.560) | -0.85 (1.662) | -1.05 (1.637) | -1.34 (1.560) | -1.07 (1.639)

48. Primary Outcome: Change From Baseline in European Quality of Life 5-Dimension (EQ-5D) Health States Visual Analog Scale (VAS) Score at Week 124
Description: as for outcome 40
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vedolizumab 300 mg (C13006 Placebo) | Vedolizumab 300 mg (C13006 Vedolizumab Q8W) | Vedolizumab 300 mg (C13006 Vedolizumab Q4W) | Vedolizumab 300 mg (C13007 Placebo) | Vedolizumab 300 mg (C13007 Vedolizumab Q8W) | Vedolizumab 300 mg (C13007 Vedolizumab Q4W) | Vedolizumab 300 mg (C13011 Placebo) | Vedolizumab 300 mg (C13011 Vedolizumab) | Vedolizumab 300 mg (C13008 De Novo Participants - UC) | Vedolizumab 300 mg (C13008 De Novo Participants - CD)
Number analyzed (Participants) | 27 | 58 | 54 | 42 | 47 | 47 | 79 | 82 | 96 | 95
score on a scale
  Baseline | 61.2 (21.60) | 61.6 (16.98) | 52.0 (16.58) | 50.0 (16.87) | 54.8 (17.87) | 52.4 (19.58) | 51.8 (16.77) | 52.8 (19.62) | 56.1 (20.59) | 55.6 (15.81)
  Change at Week 124 | 24.0 (25.45) | 19.7 (18.12) | 23.8 (21.39) | 29.4 (21.15) | 28.1 (20.71) | 24.5 (28.36) | 21.1 (21.77) | 23.8 (21.41) | 22.2 (26.13) | 18.1 (24.00)

49. Primary Outcome: Change From Baseline in European Quality of Life 5-Dimension (EQ-5D) Health States Composite Score at Week 148
Description: as for outcome 39
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vedolizumab 300 mg (C13006 Placebo) | Vedolizumab 300 mg (C13006 Vedolizumab Q8W) | Vedolizumab 300 mg (C13006 Vedolizumab Q4W) | Vedolizumab 300 mg (C13007 Placebo) | Vedolizumab 300 mg (C13007 Vedolizumab Q8W) | Vedolizumab 300 mg (C13007 Vedolizumab Q4W) | Vedolizumab 300 mg (C13011 Placebo) | Vedolizumab 300 mg (C13011 Vedolizumab) | Vedolizumab 300 mg (C13008 De Novo Participants - UC) | Vedolizumab 300 mg (C13008 De Novo Participants - CD)
Number analyzed (Participants) | 27 | 54 | 53 | 41 | 43 | 46 | 76 | 83 | 94 | 93
score on a scale
  Baseline | 7.33 (1.271) | 7.20 (1.337) | 7.64 (1.415) | 8.17 (1.447) | 7.60 (1.450) | 7.65 (1.370) | 7.75 (1.434) | 7.72 (1.541) | 7.31 (1.376) | 7.52 (1.396)
  Change at Week 148 | -1.30 (1.589) | -1.26 (1.544) | -1.62 (1.417) | -1.66 (1.559) | -1.74 (1.774) | -1.67 (1.175) | -1.11 (1.740) | -1.36 (1.679) | -1.47 (1.591) | -1.24 (1.644)

50. Primary Outcome: Change From Baseline in European Quality of Life 5-Dimension (EQ-5D) Health States Visual Analog Scale (VAS) Score at Week 148
Description: as for outcome 40
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vedolizumab 300 mg (C13006 Placebo) | Vedolizumab 300 mg (C13006 Vedolizumab Q8W) | Vedolizumab 300 mg (C13006 Vedolizumab Q4W) | Vedolizumab 300 mg (C13007 Placebo) | Vedolizumab 300 mg (C13007 Vedolizumab Q8W) | Vedolizumab 300 mg (C13007 Vedolizumab Q4W) | Vedolizumab 300 mg (C13011 Placebo) | Vedolizumab 300 mg (C13011 Vedolizumab) | Vedolizumab 300 mg (C13008 De Novo Participants - UC) | Vedolizumab 300 mg (C13008 De Novo Participants - CD)
Number analyzed (Participants) | 27 | 54 | 53 | 40 | 43 | 45 | 75 | 83 | 92 | 91
score on a scale
  Baseline | 61.2 (21.60) | 61.5 (17.24) | 51.4 (16.62) | 49.4 (17.04) | 54.3 (18.04) | 52.1 (19.63) | 51.5 (16.66) | 52.0 (19.73) | 56.2 (20.93) | 55.6 (16.31)
  Change at Week 148 | 23.4 (27.31) | 21.9 (18.53) | 28.7 (19.43) | 28.2 (20.56) | 28.2 (21.30) | 24.7 (22.11) | 24.9 (25.63) | 24.6 (22.24) | 23.9 (23.40) | 21.1 (22.50)

51. Primary Outcome: Change From Baseline in European Quality of Life 5-Dimension (EQ-5D) Health States Composite Score at Week 172
Description: as for outcome 39
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vedolizumab 300 mg (C13006 Placebo) | Vedolizumab 300 mg (C13006 Vedolizumab Q8W) | Vedolizumab 300 mg (C13006 Vedolizumab Q4W) | Vedolizumab 300 mg (C13007 Placebo) | Vedolizumab 300 mg (C13007 Vedolizumab Q8W) | Vedolizumab 300 mg (C13007 Vedolizumab Q4W) | Vedolizumab 300 mg (C13011 Placebo) | Vedolizumab 300 mg (C13011 Vedolizumab) | Vedolizumab 300 mg (C13008 De Novo Participants - UC) | Vedolizumab 300 mg (C13008 De Novo Participants - CD)
Number analyzed (Participants) | 25 | 53 | 49 | 38 | 43 | 43 | 70 | 75 | 91 | 81
score on a scale
  Baseline | 7.28 (1.308) | 7.17 (1.326) | 7.67 (1.449) | 8.03 (1.385) | 7.65 (1.446) | 7.70 (1.337) | 7.71 (1.436) | 7.81 (1.548) | 7.33 (1.407) | 7.62 (1.428)
  Change at Week 172 | -1.24 (1.535) | -1.19 (1.665) | -1.45 (1.569) | -1.76 (1.747) | -1.74 (1.747) | -1.72 (1.098) | -1.07 (1.722) | -1.27 (1.695) | -1.52 (1.546) | -1.23 (1.653)

52. Primary Outcome: Change From Baseline in European Quality of Life 5-Dimension (EQ-5D) Health States Visual Analog Scale (VAS) Score at Week 172
Description: as for outcome 40
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vedolizumab 300 mg (C13006 Placebo) | Vedolizumab 300 mg (C13006 Vedolizumab Q8W) | Vedolizumab 300 mg (C13006 Vedolizumab Q4W) | Vedolizumab 300 mg (C13007 Placebo) | Vedolizumab 300 mg (C13007 Vedolizumab Q8W) | Vedolizumab 300 mg (C13007 Vedolizumab Q4W) | Vedolizumab 300 mg (C13011 Placebo) | Vedolizumab 300 mg (C13011 Vedolizumab) | Vedolizumab 300 mg (C13008 De Novo Participants - UC) | Vedolizumab 300 mg (C13008 De Novo Participants - CD)
Number analyzed (Participants) | 25 | 53 | 48 | 38 | 43 | 42 | 70 | 75 | 90 | 80
score on a scale
  Baseline | 61.6 (22.40) | 62.1 (16.84) | 51.3 (16.87) | 49.7 (17.87) | 54.2 (17.79) | 52.4 (20.42) | 51.3 (16.58) | 50.9 (19.40) | 55.9 (20.95) | 55.4 (15.90)
  Change at Week 172 | 19.8 (27.91) | 20.3 (21.59) | 25.9 (21.53) | 29.2 (22.92) | 29.4 (21.40) | 25.9 (25.70) | 26.0 (20.30) | 23.9 (23.72) | 25.2 (22.04) | 22.2 (21.21)

53. Primary Outcome: Change From Baseline in European Quality of Life 5-Dimension (EQ-5D) Health States Composite Score at Week 196
Description: as for outcome 39
Time Frame: as for outcome 13
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vedolizumab 300 mg (C13006 Placebo) | Vedolizumab 300 mg (C13006 Vedolizumab Q8W) | Vedolizumab 300 mg (C13006 Vedolizumab Q4W) | Vedolizumab 300 mg (C13007 Placebo) | Vedolizumab 300 mg (C13007 Vedolizumab Q8W) | Vedolizumab 300 mg (C13007 Vedolizumab Q4W) | Vedolizumab 300 mg (C13011 Placebo) | Vedolizumab 300 mg (C13011 Vedolizumab) | Vedolizumab 300 mg (C13008 De Novo Participants - UC) | Vedolizumab 300 mg (C13008 De Novo Participants - CD)
Number analyzed (Participants) | 27 | 50 | 46 | 37 | 41 | 41 | 66 | 71 | 62 | 51
score on a scale
  Baseline | 7.33 (1.271) | 7.14 (1.325) | 7.54 (1.312) | 8.11 (1.487) | 7.68 (1.474) | 7.66 (1.389) | 7.71 (1.476) | 7.82 (1.579) | 7.34 (1.292) | 7.61 (1.297)
  Change at Week 196 | -1.30 (1.436) | -1.06 (1.490) | -1.52 (1.426) | -1.89 (1.449) | -1.85 (1.783) | -1.90 (1.375) | -1.12 (1.687) | -1.42 (1.555) | -1.44 (1.656) | -1.37 (1.697)

54. Primary Outcome: Change From Baseline in European Quality of Life 5-Dimension (EQ-5D) Health States Visual Analog Scale (VAS) Score at Week 196
Description: as for outcome 40
Time Frame: as for outcome 13
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vedolizumab 300 mg (C13006 Placebo) | Vedolizumab 300 mg (C13006 Vedolizumab Q8W) | Vedolizumab 300 mg (C13006 Vedolizumab Q4W) | Vedolizumab 300 mg (C13007 Placebo) | Vedolizumab 300 mg (C13007 Vedolizumab Q8W) | Vedolizumab 300 mg (C13007 Vedolizumab Q4W) | Vedolizumab 300 mg (C13011 Placebo) | Vedolizumab 300 mg (C13011 Vedolizumab) | Vedolizumab 300 mg (C13008 De Novo Participants - UC) | Vedolizumab 300 mg (C13008 De Novo Participants - CD)
Number analyzed (Participants) | 27 | 50 | 46 | 37 | 41 | 41 | 66 | 71 | 62 | 51
score on a scale
  Baseline | 61.2 (21.60) | 61.3 (16.63) | 52.5 (17.01) | 49.0 (18.41) | 54.2 (17.71) | 52.8 (20.56) | 51.5 (16.72) | 51.5 (19.58) | 56.7 (20.21) | 56.5 (14.35)
  Change at Week 196 | 22.9 (28.01) | 21.6 (17.20) | 26.4 (20.17) | 31.9 (23.39) | 29.1 (22.45) | 29.2 (22.32) | 24.6 (21.32) | 23.3 (26.17) | 22.1 (22.91) | 23.2 (18.14)

55. Primary Outcome: Change From Baseline in European Quality of Life 5-Dimension (EQ-5D) Health States Composite Score at Week 248
Description: as for outcome 39
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vedolizumab 300 mg (C13006 Placebo) | Vedolizumab 300 mg (C13006 Vedolizumab Q8W) | Vedolizumab 300 mg (C13006 Vedolizumab Q4W) | Vedolizumab 300 mg (C13007 Placebo) | Vedolizumab 300 mg (C13007 Vedolizumab Q8W) | Vedolizumab 300 mg (C13007 Vedolizumab Q4W) | Vedolizumab 300 mg (C13011 Placebo) | Vedolizumab 300 mg (C13011 Vedolizumab) | Vedolizumab 300 mg (C13008 De Novo Participants - UC) | Vedolizumab 300 mg (C13008 De Novo Participants - CD)
Number analyzed (Participants) | 21 | 38 | 36 | 32 | 32 | 31 | 38 | 45 | 3 | 4
score on a scale
  Baseline | 7.48 (1.365) | 7.21 (1.119) | 7.69 (1.215) | 8.09 (1.510) | 7.66 (1.450) | 7.84 (1.463) | 7.63 (1.532) | 7.89 (1.541) | 7.33 (1.155) | 7.75 (1.500)
  Change at Week 248 | -1.67 (1.653) | -1.03 (1.619) | -1.58 (1.339) | -2.03 (1.425) | -1.81 (1.554) | -1.97 (1.538) | -1.05 (2.039) | -1.57 (1.521) | -2.00 (1.000) | -2.00 (1.414)

56. Primary Outcome: Change From Baseline in European Quality of Life 5-Dimension (EQ-5D) Health States Visual Analog Scale (VAS) Score at Week 248
Description: as for outcome 40
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vedolizumab 300 mg (C13006 Placebo) | Vedolizumab 300 mg (C13006 Vedolizumab Q8W) | Vedolizumab 300 mg (C13006 Vedolizumab Q4W) | Vedolizumab 300 mg (C13007 Placebo) | Vedolizumab 300 mg (C13007 Vedolizumab Q8W) | Vedolizumab 300 mg (C13007 Vedolizumab Q4W) | Vedolizumab 300 mg (C13011 Placebo) | Vedolizumab 300 mg (C13011 Vedolizumab) | Vedolizumab 300 mg (C13008 De Novo Participants - UC) | Vedolizumab 300 mg (C13008 De Novo Participants - CD)
Number analyzed (Participants) | 21 | 37 | 36 | 32 | 32 | 31 | 38 | 45 | 3 | 4
score on a scale
  Baseline | 57.2 (21.28) | 61.6 (16.17) | 52.1 (16.63) | 47.2 (18.17) | 52.3 (16.40) | 53.2 (19.72) | 50.8 (17.39) | 49.0 (19.37) | 61.3 (28.11) | 47.5 (7.33)
  Change at Week 248 | 27.5 (25.77) | 17.7 (18.62) | 28.0 (22.14) | 34.9 (18.79) | 32.1 (19.98) | 29.9 (24.37) | 24.7 (25.34) | 28.9 (27.65) | 28.7 (32.72) | 34.3 (11.44)

57. Primary Outcome: Change From Baseline in European Quality of Life 5-Dimension (EQ-5D) Health States Composite Score at Week 300
Description: as for outcome 39
Time Frame: as for outcome 15
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vedolizumab 300 mg (C13006 Placebo) | Vedolizumab 300 mg (C13006 Vedolizumab Q8W) | Vedolizumab 300 mg (C13006 Vedolizumab Q4W) | Vedolizumab 300 mg (C13007 Placebo) | Vedolizumab 300 mg (C13007 Vedolizumab Q8W) | Vedolizumab 300 mg (C13007 Vedolizumab Q4W) | Vedolizumab 300 mg (C13011 Placebo) | Vedolizumab 300 mg (C13011 Vedolizumab)
Number analyzed (Participants) | 7 | 14 | 13 | 9 | 8 | 16 | 4 | 2
score on a scale
  Baseline | 8.14 (1.069) | 7.50 (0.941) | 8.08 (1.115) | 8.33 (1.803) | 7.88 (1.356) | 7.94 (1.063) | 7.75 (2.062) | 7.00 (0.000)
  Change at Week 300 | -2.29 (1.799) | -1.43 (2.065) | -1.77 (1.363) | -2.11 (1.965) | -2.00 (2.138) | -2.25 (1.438) | -1.50 (1.291) | 0.50 (2.121)

58. Primary Outcome: Change From Baseline in EuroQol 5D Health States (EQ-5D) Visual Analog Scale (VAS) Score at Week 300
Description: as for outcome 40
Time Frame: as for outcome 15
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vedolizumab 300 mg (C13006 Placebo) | Vedolizumab 300 mg (C13006 Vedolizumab Q8W) | Vedolizumab 300 mg (C13006 Vedolizumab Q4W) | Vedolizumab 300 mg (C13007 Placebo) | Vedolizumab 300 mg (C13007 Vedolizumab Q8W) | Vedolizumab 300 mg (C13007 Vedolizumab Q4W) | Vedolizumab 300 mg (C13011 Placebo) | Vedolizumab 300 mg (C13011 Vedolizumab)
Number analyzed (Participants) | 7 | 14 | 13 | 9 | 8 | 16 | 4 | 2
score on a scale
  Baseline | 58.1 (20.27) | 64.9 (11.82) | 55.7 (10.10) | 50.4 (22.34) | 53.1 (15.80) | 42.9 (19.54) | 43.5 (19.12) | 52.0 (24.04)
  Change at Week 300 | 23.6 (29.14) | 20.4 (17.92) | 28.4 (14.78) | 33.2 (25.83) | 31.3 (17.47) | 43.6 (23.17) | 40.3 (9.50) | 13.0 (11.31)

59. Primary Outcome: Change From Baseline in European Quality of Life 5-Dimension (EQ-5D) Health States Composite Score at Week 352
Description: as for outcome 39
Time Frame: as for outcome 16
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vedolizumab 300 mg (C13006 Placebo) | Vedolizumab 300 mg (C13006 Vedolizumab Q8W) | Vedolizumab 300 mg (C13006 Vedolizumab Q4W) | Vedolizumab 300 mg (C13007 Placebo) | Vedolizumab 300 mg (C13007 Vedolizumab Q8W) | Vedolizumab 300 mg (C13007 Vedolizumab Q4W)
Number analyzed (Participants) | 1 | 1 | 3 | 1 | 2 | 1
score on a scale
  Baseline | 8.00 (NA) — SD was not calculated for 1 participant. | 8.00 (NA) — SD was not calculated for 1 participant. | 8.33 (0.577) | 12.00 (NA) — SD was not calculated for 1 participant. | 8.00 (1.414) | 9.00 (NA) — SD was not calculated for 1 participant.
  Change at Week 352 | -2.00 (NA) — SD was not calculated for 1 participant. | -3.00 (NA) — SD was not calculated for 1 participant. | -1.33 (1.528) | -6.00 (NA) — SD was not calculated for 1 participant. | -1.00 (0.000) | -4.00 (NA) — SD was not calculated for 1 participant.

60. Primary Outcome: Change From Baseline in European Quality of Life 5-Dimension (EQ-5D) Health States Visual Analog Scale (VAS) Score at Week 352
Description: as for outcome 40
Time Frame: as for outcome 16
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vedolizumab 300 mg (C13006 Placebo) | Vedolizumab 300 mg (C13006 Vedolizumab Q8W) | Vedolizumab 300 mg (C13006 Vedolizumab Q4W) | Vedolizumab 300 mg (C13007 Placebo) | Vedolizumab 300 mg (C13007 Vedolizumab Q8W) | Vedolizumab 300 mg (C13007 Vedolizumab Q4W)
Number analyzed (Participants) | 1 | 1 | 3 | 1 | 2 | 1
score on a scale
  Baseline | 52.0 (NA) — SD was not calculated for 1 participant. | 50.0 (NA) — SD was not calculated for 1 participant. | 48.0 (8.19) | 15.0 (NA) — SD was not calculated for 1 participant. | 50.0 (14.14) | 31.0 (NA) — SD was not calculated for 1 participant.
  Change at Week 352 | 46.0 (NA) — SD was not calculated for 1 participant. | 40.0 (NA) — SD was not calculated for 1 participant. | 24.3 (20.11) | 64.0 (NA) — SD was not calculated for 1 participant. | 24.0 (8.49) | 59.0 (NA) — SD was not calculated for 1 participant.

ADVERSE EVENTS:
Time Frame: From first dose of study drug in this study through 16 weeks after the last dose of study drug (Up to approximately 8.5 years)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Groups:
- Vedolizumab 300 mg: Vedolizumab 300 mg, 30-minute IV infusion, Q4W, up to approximately 260 weeks. Includes De Novo participants and participants previously enrolled in studies C13004, C13006, C13007 and C13011.
Arm/Group | Vedolizumab 300 mg
All-Cause Mortality (participants affected / at risk) | 10/2243
Serious Adverse Events (participants affected / at risk) | 825/2243
Other Adverse Events (participants affected / at risk) | 1820/2243
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vedolizumab 300 mg (N=2243)
Crohn's disease (Gastrointestinal disorders) | 225
Enteritis (Gastrointestinal disorders) | 1
Epiploic appendagitis (Gastrointestinal disorders) | 1
Gastrointestinal inflammation (Gastrointestinal disorders) | 2
Pouchitis (Gastrointestinal disorders) | 1
Colitis ulcerative (Gastrointestinal disorders) | 120
Colitis (Gastrointestinal disorders) | 3
Colitis ischaemic (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 50
Abdominal pain upper (Gastrointestinal disorders) | 6
Abdominal pain lower (Gastrointestinal disorders) | 2
Small intestinal obstruction (Gastrointestinal disorders) | 29
Ileal stenosis (Gastrointestinal disorders) | 14
Small intestinal stenosis (Gastrointestinal disorders) | 2
Intestinal obstruction (Gastrointestinal disorders) | 17
Intestinal stenosis (Gastrointestinal disorders) | 6
Ileus (Gastrointestinal disorders) | 8
Subileus (Gastrointestinal disorders) | 5
Anal fistula (Gastrointestinal disorders) | 15
Enterocolonic fistula (Gastrointestinal disorders) | 2
Enterocutaneous fistula (Gastrointestinal disorders) | 2
Enterovesical fistula (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 10
Nausea (Gastrointestinal disorders) | 7
Diarrhoea (Gastrointestinal disorders) | 9
Rectal haemorrhage (Gastrointestinal disorders) | 6
Intestinal haemorrhage (Gastrointestinal disorders) | 1
Colonic stenosis (Gastrointestinal disorders) | 5
Colonic obstruction (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 4
Haematochezia (Gastrointestinal disorders) | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 5
Pancreatitis acute (Gastrointestinal disorders) | 1
Large intestine perforation (Gastrointestinal disorders) | 5
Intestinal perforation (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 6
Constipation (Gastrointestinal disorders) | 4
Colon dysplasia (Gastrointestinal disorders) | 3
Inguinal hernia (Gastrointestinal disorders) | 3
Abdominal hernia (Gastrointestinal disorders) | 4
Abdominal hernia obstructive (Gastrointestinal disorders) | 2
Anal stenosis (Gastrointestinal disorders) | 1
Rectal stenosis (Gastrointestinal disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 2
Food poisoning (Gastrointestinal disorders) | 2
Haemorrhoids (Gastrointestinal disorders) | 2
Peritonitis (Gastrointestinal disorders) | 2
Mouth ulceration (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Anal fissure (Gastrointestinal disorders) | 1
Proctalgia (Gastrointestinal disorders) | 1
Duodenal ulcer (Gastrointestinal disorders) | 1
Intestinal ischaemia (Gastrointestinal disorders) | 1
Megacolon (Gastrointestinal disorders) | 1
Periproctitis (Gastrointestinal disorders) | 1
Umbilical hernia (Gastrointestinal disorders) | 1
Anal abscess (Infections and infestations) | 33
Gastroenteritis (Infections and infestations) | 19
Appendicitis (Infections and infestations) | 17
Abdominal abscess (Infections and infestations) | 13
Perirectal abscess (Infections and infestations) | 4
Diverticulitis (Infections and infestations) | 3
Diarrhoea infectious (Infections and infestations) | 3
Abdominal wall abscess (Infections and infestations) | 1
Appendicitis perforated (Infections and infestations) | 2
Enterocolitis infectious (Infections and infestations) | 1
Gastrointestinal infection (Infections and infestations) | 1
Rectal abscess (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 21 — One treatment-emergent death occurred during treatment with vedolizumab 300 mg and is not related.
Lobar pneumonia (Infections and infestations) | 2
Bronchitis (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Clostridium difficile colitis (Infections and infestations) | 11
Clostridial infection (Infections and infestations) | 5
Clostridium colitis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 7
Arthritis bacterial (Infections and infestations) | 1
Asymptomatic bacteriuria (Infections and infestations) | 1
Vaginal cellulitis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 6 — One treatment-emergent death occurred during treatment with vedolizumab 300 mg and was not related.
Septic shock (Infections and infestations) | 3
Abdominal sepsis (Infections and infestations) | 2
Urosepsis (Infections and infestations) | 1
Gastroenteritis viral (Infections and infestations) | 3
Meningitis viral (Infections and infestations) | 2
Viral infection (Infections and infestations) | 4
Pneumonia viral (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 2
Laryngitis (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Peritonsillar abscess (Infections and infestations) | 2
Tonsillitis (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 1
Pelvic abscess (Infections and infestations) | 4
Abscess (Infections and infestations) | 1
Postoperative wound infection (Infections and infestations) | 2
Subcutaneous abscess (Infections and infestations) | 2
Blister infected (Infections and infestations) | 1
Pilonidal cyst (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 5
Cytomegalovirus colitis (Infections and infestations) | 3
Pulmonary tuberculosis (Infections and infestations) | 3
Oesophageal candidiasis (Infections and infestations) | 1
Vulvovaginal candidiasis (Infections and infestations) | 1
Influenza (Infections and infestations) | 2
Klebsiella infection (Infections and infestations) | 1
Klebsiella sepsis (Infections and infestations) | 1
Abscess jaw (Infections and infestations) | 1
Campylobacter intestinal infection (Infections and infestations) | 1
Meningitis (Infections and infestations) | 1
Cryptosporidiosis infection (Infections and infestations) | 1
Tooth abscess (Infections and infestations) | 1
Infectious mononucleosis (Infections and infestations) | 1
Vulval abscess (Infections and infestations) | 1
West Nile viral infection (Infections and infestations) | 1 — One treatment-emergent death occurred during treatment with vedolizumab 300 mg and was related.
Giardiasis (Infections and infestations) | 1
Cholangitis suppurative (Infections and infestations) | 1
Herpes simplex (Infections and infestations) | 1
Psoas abscess (Infections and infestations) | 1
Gastroenteritis salmonella (Infections and infestations) | 2
Tinea pedis (Infections and infestations) | 1
Infusion site infection (Infections and infestations) | 1
Intestinal anastomosis complication (Injury, poisoning and procedural complications) | 6
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 4
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 2
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 2
Postoperative ileus (Injury, poisoning and procedural complications) | 1
Humerus fracture (Injury, poisoning and procedural complications) | 4
Hand fracture (Injury, poisoning and procedural complications) | 3
Ulna fracture (Injury, poisoning and procedural complications) | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1
Femur fracture (Injury, poisoning and procedural complications) | 3
Ankle fracture (Injury, poisoning and procedural complications) | 2
Anastomotic stenosis (Injury, poisoning and procedural complications) | 1
Incisional hernia (Injury, poisoning and procedural complications) | 3
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2
Procedural site reaction (Injury, poisoning and procedural complications) | 2
Infusion related reaction (Injury, poisoning and procedural complications) | 1
Post procedural discharge (Injury, poisoning and procedural complications) | 1
Procedural pain (Injury, poisoning and procedural complications) | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1
Fibula fracture (Injury, poisoning and procedural complications) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Joint injury (Injury, poisoning and procedural complications) | 2
Meniscus lesion (Injury, poisoning and procedural complications) | 2
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 2
Traumatic lung injury (Injury, poisoning and procedural complications) | 1
Dislocation of vertebra (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1
Intentional overdose (Injury, poisoning and procedural complications) | 1
Overdose (Injury, poisoning and procedural complications) | 2
Acetabulum fracture (Injury, poisoning and procedural complications) | 1
Pubis fracture (Injury, poisoning and procedural complications) | 1
Accidental poisoning (Injury, poisoning and procedural complications) | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 1
Rib fracture (Injury, poisoning and procedural complications) | 2
Splenic rupture (Injury, poisoning and procedural complications) | 1
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1 — One treatment-emergent death occurred during treatment with vedolizumab 300 mg and was not related.
Joint dislocation (Injury, poisoning and procedural complications) | 1
Tendon injury (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Urethral injury (Injury, poisoning and procedural complications) | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Carcinoid tumour of the appendix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 — One treatment-emergent death occurred during treatment with vedolizumab 300 mg and was related.
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 — One treatment-emergent death occurred during treatment with vedolizumab 300 mg and is not related.
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Spinal meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neurilemmoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 5
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Joint effusion (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 5
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Fistula (Musculoskeletal and connective tissue disorders) | 1
Fistula discharge (Musculoskeletal and connective tissue disorders) | 1
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 1
Spondyloarthropathy (Musculoskeletal and connective tissue disorders) | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 2
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 2
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Muscle disorder (Musculoskeletal and connective tissue disorders) | 1
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 7
Cholecystitis (Hepatobiliary disorders) | 7
Cholecystitis acute (Hepatobiliary disorders) | 5
Cholecystitis chronic (Hepatobiliary disorders) | 1
Biliary colic (Hepatobiliary disorders) | 2
Cholangitis (Hepatobiliary disorders) | 2
Cholangitis sclerosing (Hepatobiliary disorders) | 2
Bile duct stone (Hepatobiliary disorders) | 4
Jaundice (Hepatobiliary disorders) | 1
Hepatitis acute (Hepatobiliary disorders) | 1
Non-cardiac chest pain (General disorders) | 7
Chest discomfort (General disorders) | 1
Chest pain (General disorders) | 1
Pain (General disorders) | 1
Asthenia (General disorders) | 3
Fatigue (General disorders) | 3
Pyrexia (General disorders) | 4
Hernia obstructive (General disorders) | 2
Device dislocation (General disorders) | 1
Influenza like illness (General disorders) | 1
Pseudopolyp (General disorders) | 1
No therapeutic response (General disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 10 — One treatment-emergent death occurred during treatment with vedolizumab 300 mg and was not related.
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 4
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4
Asthma (Respiratory, thoracic and mediastinal disorders) | 2
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 — One treatment-emergent death occurred during treatment with vedolizumab 300 mg and was not related.
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 3 — One treatment-emergent death occurred during treatment with vedolizumab 300 mg and was not related.
Subarachnoid haemorrhage (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 4
Lumbar radiculopathy (Nervous system disorders) | 1
Sciatica (Nervous system disorders) | 1
Intracranial aneurysm (Nervous system disorders) | 1
Carotid artery stenosis (Nervous system disorders) | 3
Aphasia (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
VIIth nerve paralysis (Nervous system disorders) | 1
Grand mal convulsion (Nervous system disorders) | 1
Headache (Nervous system disorders) | 4
Transient global amnesia (Nervous system disorders) | 1
Migraine (Nervous system disorders) | 1
Carpal tunnel syndrome (Nervous system disorders) | 1
Multiple sclerosis (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Optic neuritis (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Convulsion (Nervous system disorders) | 2
Hypoaesthesia (Nervous system disorders) | 1
Spinal cord compression (Nervous system disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 11
Calculus urinary (Renal and urinary disorders) | 1
Renal colic (Renal and urinary disorders) | 4
Dysuria (Renal and urinary disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 1
Bladder hypertrophy (Renal and urinary disorders) | 1
Bladder prolapse (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 2
Ureteric stenosis (Renal and urinary disorders) | 1
Urethral prolapse (Renal and urinary disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 14
Iron deficiency anaemia (Blood and lymphatic system disorders) | 5
Febrile neutropenia (Blood and lymphatic system disorders) | 3
Pancytopenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 6
Hypokalaemia (Metabolism and nutrition disorders) | 5
Malnutrition (Metabolism and nutrition disorders) | 3
Obesity (Metabolism and nutrition disorders) | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1
Hypoproteinaemia (Metabolism and nutrition disorders) | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Iron deficiency (Metabolism and nutrition disorders) | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 5
Metrorrhagia (Reproductive system and breast disorders) | 1
Cervical dysplasia (Reproductive system and breast disorders) | 2
Uterine cervical erosion (Reproductive system and breast disorders) | 1
Menorrhagia (Reproductive system and breast disorders) | 2
Ovarian adhesion (Reproductive system and breast disorders) | 1
Ovarian mass (Reproductive system and breast disorders) | 1
Female genital tract fistula (Reproductive system and breast disorders) | 3
Breast haematoma (Reproductive system and breast disorders) | 1
Cystocele (Reproductive system and breast disorders) | 1
Uterine polyp (Reproductive system and breast disorders) | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1
Myocardial infarction (Cardiac disorders) | 3
Myocardial ischaemia (Cardiac disorders) | 2
Angina pectoris (Cardiac disorders) | 2
Atrial fibrillation (Cardiac disorders) | 4
Supraventricular tachycardia (Cardiac disorders) | 2
Myopericarditis (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 1
Pericarditis (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Ventricular tachycardia (Cardiac disorders) | 1
Depression (Psychiatric disorders) | 4
Stress (Psychiatric disorders) | 2
Anxiety (Psychiatric disorders) | 1
Mental status changes (Psychiatric disorders) | 3
Homicidal ideation (Psychiatric disorders) | 1
Affective disorder (Psychiatric disorders) | 1
Alcohol abuse (Psychiatric disorders) | 1
Completed suicide (Psychiatric disorders) | 1 — One treatment-emergent death occurred during treatment with vedolizumab 300 mg and was not related.
Deep vein thrombosis (Vascular disorders) | 3
Axillary vein thrombosis (Vascular disorders) | 1
Subclavian vein thrombosis (Vascular disorders) | 1
Thrombophlebitis superficial (Vascular disorders) | 1
Hypertension (Vascular disorders) | 2
Thrombosis (Vascular disorders) | 1
Arteriosclerosis (Vascular disorders) | 1
Varicose vein (Vascular disorders) | 1
Weight decreased (Investigations) | 2
Blood glucose increased (Investigations) | 1
Hepatic enzyme increased (Investigations) | 1
C-reactive protein increased (Investigations) | 1
Haemoglobin decreased (Investigations) | 1
Blood creatinine increased (Investigations) | 1
Rash (Skin and subcutaneous tissue disorders) | 2
Systemic lupus erythematosus rash (Skin and subcutaneous tissue disorders) | 1
Pyoderma gangrenosum (Skin and subcutaneous tissue disorders) | 2
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 1
Scar (Skin and subcutaneous tissue disorders) | 1
Uveitis (Eye disorders) | 2
Cataract (Eye disorders) | 1
Vitreous floaters (Eye disorders) | 1
Retinal detachment (Eye disorders) | 1
Vision blurred (Eye disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Vertigo positional (Ear and labyrinth disorders) | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1
Vitello-intestinal duct remnant (Congenital, familial and genetic disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1
Calculus ureteric (Renal and urinary disorders) | 4
Malaise (General disorders) | 2
General physical health deterioration (General disorders) | 1
Renal failure acute (Renal and urinary disorders) | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 1
Skeletal injury (Injury, poisoning and procedural complications) | 1
Thermal burn (Injury, poisoning and procedural complications) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Chondropathy (Musculoskeletal and connective tissue disorders) | 1
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Cervicobrachial syndrome (Nervous system disorders) | 1
Intracranial hypotension (Nervous system disorders) | 1
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Spinal cord neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 1
Prostatitis (Reproductive system and breast disorders) | 1
Arteriospasm coronary (Cardiac disorders) | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 1
Psychotic disorder (Psychiatric disorders) | 1
Peripheral vascular disorder (Vascular disorders) | 1
Peripheral ischaemia (Vascular disorders) | 1
Femoral arterial stenosis (Vascular disorders) | 1
Liver function test abnormal (Investigations) | 1
Lymphocyte count decreased (Investigations) | 1
Serum sickness (Immune system disorders) | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Intestinal fistula (Gastrointestinal disorders) | 1
Rectourethral fistula (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 1
Small intestinal perforation (Gastrointestinal disorders) | 1
Inguinal hernia strangulated (Gastrointestinal disorders) | 1
Anal inflammation (Gastrointestinal disorders) | 1
Faecaloma (Gastrointestinal disorders) | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 1
Umbilical hernia, obstructive (Gastrointestinal disorders) | 1
Vulval cellulitis (Infections and infestations) | 1
Enterocolitis viral (Infections and infestations) | 1
Vestibular neuronitis (Infections and infestations) | 1
Acute sinusitis (Infections and infestations) | 1
Postoperative abscess (Infections and infestations) | 2
Incision site infection (Infections and infestations) | 1
Peridiverticular abscess (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Pyelonephritis acute (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Herpes zoster ophthalmic (Infections and infestations) | 1
Ear infection (Infections and infestations) | 1
Mastoiditis (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vedolizumab 300 mg (N=2243)
Nasopharyngitis (Infections and infestations) | 594
Upper respiratory tract infection (Infections and infestations) | 379
Sinusitis (Infections and infestations) | 235
Bronchitis (Infections and infestations) | 216
Gastroenteritis (Infections and infestations) | 216
Influenza (Infections and infestations) | 208
Urinary tract infection (Infections and infestations) | 175
Abdominal pain (Gastrointestinal disorders) | 393
Crohn's disease (Gastrointestinal disorders) | 333
Nausea (Gastrointestinal disorders) | 333
Diarrhoea (Gastrointestinal disorders) | 284
Colitis ulcerative (Gastrointestinal disorders) | 251
Vomiting (Gastrointestinal disorders) | 227
Abdominal pain upper (Gastrointestinal disorders) | 139
Arthralgia (Musculoskeletal and connective tissue disorders) | 482
Back pain (Musculoskeletal and connective tissue disorders) | 239
Pain in extremity (Musculoskeletal and connective tissue disorders) | 125
Myalgia (Musculoskeletal and connective tissue disorders) | 121
Headache (Nervous system disorders) | 452
Dizziness (Nervous system disorders) | 162
Pyrexia (General disorders) | 277
Fatigue (General disorders) | 229
Influenza like illness (General disorders) | 148
Cough (Respiratory, thoracic and mediastinal disorders) | 251
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 168
Anaemia (Blood and lymphatic system disorders) | 181
Rash (Skin and subcutaneous tissue disorders) | 153
Insomnia (Psychiatric disorders) | 122

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In general, Investigators may publish clinical data after the earlier of (i) publication by the Sponsor or (ii) 12 months following the abandonment, early termination or database lock; provided a copy of the publication provided to Sponsor at least 30 days ahead of publication, the Sponsor's confidential information is removed as may be requested by Sponsor and Investigator defers publication for up to 60 days in the event Sponsor provides notice that it intends to file a patent application.

DOCUMENTS (2):
  • Study Protocol (2016-08-22): https://cdn.clinicaltrials.gov/large-docs/33/NCT00790933/Prot_001.pdf
  • Statistical Analysis Plan (2013-01-07): https://cdn.clinicaltrials.gov/large-docs/33/NCT00790933/SAP_000.pdf